CLINICAL TRIAL: NCT03529773
Title: A PHASE 1/2, PLACEBO-CONTROLLED, RANDOMIZED, OBSERVER-BLIND, DOSE-FINDING, FIRST-IN-HUMAN STUDY TO DESCRIBE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A RESPIRATORY SYNCYTIAL VIRUS (RSV) VACCINE IN HEALTHY ADULTS
Brief Title: A Study to Describe the Safety and Immunogenicity of a RSV Vaccine in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C3671001; RSV FIH (Other: Alias Study Number)
Record Dates: First submitted 2018-04-17; First posted 2018-05-18 (Actual); Results first posted 2021-03-04 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Tract Infections
Keywords: Respiratory tract infections, RSV, vaccine
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (20):
- Sentinel Arm 1 (Experimental): Low dose formulation A
  Interventions: Biological: Formulation A
- Sentinel Arm 2 (Experimental): Mid dose formulation A
  Interventions: Biological: Formulation A
- Sentinel Arm 3 (Experimental): High dose formulation A
  Interventions: Biological: Formulation A
- Sentinel Arm 4 (Experimental): Low dose formulation B
  Interventions: Biological: Formulation B
- Sentinel Arm 5 (Experimental): Mid dose formulation B
  Interventions: Biological: Formulation B
- Sentinel Arm 6 (Experimental): High dose formulation B
  Interventions: Biological: Formulation B
- Sentinel Arm 7 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- Expanded Arm 8 (Experimental): Low dose formulation A and SIIV
  Interventions: Biological: Formulation A
- Expanded Arm 9 (Experimental): Mid dose formulation A and SIIV
  Interventions: Biological: Formulation A
- Expanded Arm 10 (Experimental): High dose formulation A and SIIV
  Interventions: Biological: Formulation A
- Expanded Arm 11 (Experimental): Low dose formulation B and SIIV
  Interventions: Biological: Formulation B
- Expanded Arm 12 (Experimental): Mid dose formulation B and SIIV
  Interventions: Biological: Formulation B
- Expanded Arm 13 (Experimental): High dose formulation B and SIIV
  Interventions: Biological: Formulation B
- Expanded Arm 14 (Experimental): Low dose formulation A and placebo
  Interventions: Biological: Formulation A
- Expanded Arm 15 (Experimental): Mid dose formulation A and placebo
  Interventions: Biological: Formulation A
- Expanded Arm 16 (Experimental): High dose formulation A and placebo
  Interventions: Biological: Formulation A
- Expanded Arm 17 (Experimental): Low dose formulation B and placebo
  Interventions: Biological: Formulation B
- Expanded Arm 18 (Experimental): Mid dose formulation B and placebo
  Interventions: Biological: Formulation B
- Expanded Arm 19 (Experimental): High dose formulation B and placebo
  Interventions: Biological: Formulation B
- Expanded Arm 20 (Placebo Comparator): placebo and placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Formulation A — RSV vaccine
  Arms: Expanded Arm 10; Expanded Arm 14; Expanded Arm 15; Expanded Arm 16; Expanded Arm 8; Expanded Arm 9; Sentinel Arm 1; Sentinel Arm 2; Sentinel Arm 3
Biological: Formulation B — RSV vaccine
  Arms: Expanded Arm 11; Expanded Arm 12; Expanded Arm 13; Expanded Arm 17; Expanded Arm 18; Expanded Arm 19; Sentinel Arm 4; Sentinel Arm 5; Sentinel Arm 6
Biological: Placebo — Placebo
  Arms: Expanded Arm 20; Sentinel Arm 7

SUMMARY:
The study will describe the safety, tolerability, and immunogenicity of up to 6 RSV vaccine formulations when administered alone or concomitantly with seasonal inactivated influenza vaccine (SIIV).

DETAILED DESCRIPTION:
The study will describe the safety, tolerability, and immunogenicity of up to 6 RSV vaccine formulations when administered alone or concomitantly with SIIV. Healthy male and female subjects divided into 2 age groups (18-49 years of age and 50-85 years of age in the sentinel cohort and 18-49 years of age and 65-85 years of age in the expanded cohort) will be enrolled. Age groups will run in parallel. Subjects in the sentinel cohort in each age group will receive one of two RSV vaccine formulations at one of 3 antigen dose levels or placebo. Subjects in the expanded cohort in each age group will receive one of two RSV vaccine formulations at one of 3 antigen dose levels with and without SIIV.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject has been informed of all pertinent aspects of the study.
2. Healthy adults who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
3. Willing and able to comply with scheduled visits, vaccination plan, laboratory tests, and other study procedures.
4. Male subject who is able to father children and willing to use a highly effective method of contraception as outlined in this protocol until at least 28 days after the last dose of investigational product; female subject who is of childbearing potential and at risk for pregnancy and who is willing to use a highly effective method of contraception as outlined in this protocol until at least 28 days after the last dose of investigational product; male subject not able to father children; female subject not of childbearing potential.
5. Sentinel-cohort subjects only: Male and female adults aged 18 to 85 years at the time of enrollment (signing of the ICD).
6. Expanded-cohort subjects only: Male and female adults aged 18 to 49 years of age or 65 to 85 years at the time of enrollment (signing of the ICD).

Exclusion Criteria:

1. Sentinel-cohort subjects only: Any screening hematology and/or blood chemistry laboratory value that meets the definition of a ≥ Grade 1 abnormality.
2. Sentinel-cohort subjects only: Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (HBc Abs), or hepatitis C virus antibodies (HCV Abs) at the screening visit.
3. Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
4. Participation in other studies involving investigational product within 28 days prior to study entry and/or during study participation.
5. Known infection with HIV, hepatitis C virus (HCV), or hepatitis B virus (HBV).
6. Previous vaccination with any licensed or investigational RSV vaccine, or planned receipt throughout the study of nonstudy RSV vaccine.
7. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the investigational product(s).
8. Immunocompromised subjects with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
9. Subjects who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, eg, for cancer or an autoimmune disease, or planned receipt throughout the study. If systemic corticosteroids have been administered short term (<14 days) for treatment of an acute illness, subjects should not be enrolled into the study until corticosteroid therapy has been discontinued for at least 28 days before investigational product administration. Intra-articular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
10. Subject with a history of autoimmune disease or an active autoimmune disease requiring therapeutic intervention including but not limited to: systemic or cutaneous lupus erythematosus, autoimmune arthritis/rheumatoid arthritis, Guillain-Barré syndrome, multiple sclerosis, Sjögren's syndrome, idiopathic thrombocytopenia purpura, glomerulonephritis, autoimmune thyroiditis, giant cell arteritis (temporal arteritis), psoriasis, and insulin-dependent diabetes mellitus (type 1).
11. Receipt of blood/plasma products or immunoglobulin, from 60 days before investigational product administration or planned receipt throughout the study.
12. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
13. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection.
14. Women who are pregnant or breastfeeding.
15. Expanded-cohort subjects only: Vaccination with any influenza vaccine within 6 months (182 days) before investigational product administration.
16. Expanded-cohort subjects only: Allergy to egg proteins (egg or egg products) or chicken proteins.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1235 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (40):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Anaheim Clinical Trials, Anaheim, California
  - Paradigm Clinical Research Centers, Inc., La Mesa, California
  - Paradigm Clinical Research Center, Redding, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Meridian Clinical Research Dakota Dunes, Sioux City, Iowa
  - Augusta Family Practice, Augusta, Kansas
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Axtell Clinic, P.A., Newton, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - United Medical Associates, Binghamton, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Rochester Regional Health/Rochester General Hospital, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Raleigh, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Benchmark Research, Austin, Texas
  - Texas Health Care, PLLC, Fort Worth, Texas
  - Ventavia Research Group, LLC, Fort Worth, Texas
  - Benchmark Research, Fort Worth, Texas
  - HealthFirst Medical Group, Fort Worth, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. /Foothill Family Clinic South, Salt Lake City, Utah
  - J.Lewis Research, Inc. / Jordan River Family Medicine, South Jordan, Utah
  - Advanced Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
Time Frame: Starting 24 months after study completion.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Walsh EE, Falsey AR, Zareba AM, Jiang Q, Gurtman A, Radley D, Gomme E, Cooper D, Jansen KU, Gruber WC, Swanson KA, Schmoele-Thoma B. Respiratory Syncytial Virus Prefusion F Vaccination: Antibody Persistence and Revaccination. J Infect Dis. 2024 Oct 16;230(4):e905-e916. doi: 10.1093/infdis/jiae185. PMID 38606958
- [Derived] Walsh EE, Falsey AR, Scott DA, Gurtman A, Zareba AM, Jansen KU, Gruber WC, Dormitzer PR, Swanson KA, Radley D, Gomme E, Cooper D, Schmoele-Thoma B. A Randomized Phase 1/2 Study of a Respiratory Syncytial Virus Prefusion F Vaccine. J Infect Dis. 2022 Apr 19;225(8):1357-1366. doi: 10.1093/infdis/jiab612. PMID 34932102
- [Derived] Falsey AR, Walsh EE, Scott DA, Gurtman A, Zareba A, Jansen KU, Gruber WC, Dormitzer PR, Swanson KA, Jiang Q, Gomme E, Cooper D, Schmoele-Thoma B. Phase 1/2 Randomized Study of the Immunogenicity, Safety, and Tolerability of a Respiratory Syncytial Virus Prefusion F Vaccine in Adults With Concomitant Inactivated Influenza Vaccine. J Infect Dis. 2022 Jun 15;225(12):2056-2066. doi: 10.1093/infdis/jiab611. PMID 34931667
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3671001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 1446 participants signed the Informed Consent Form (ICF). Out of which 211 participants were screen failures,1235 actually enrolled into the study and assigned to a study treatment. Only 1233 participants were vaccinated.
Groups:
- Sentinel Cohort: Respiratory Syncytial Virus (RSV) Vaccine 60 Microgram (mcg) Age 18-49 Years: Participants aged 18-49 years received single 60-mcg dose of RSV vaccine, intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years: Participants aged 18-49 years received single 60-mcg dose with aluminum hydroxide intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 120 mcg Age 18-49 Years: Participants aged 18-49 years received single 120-mcg dose intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years: Participants aged 18-49 years received single 120-mcg dose with aluminum hydroxide intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 240 mcg Age 18-49 Years: Participants aged 18-49 years received single 240-mcg dose intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years: Participants aged 18-49 years received single 240-mcg dose with aluminum hydroxide intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: Placebo Age 18-49 Years: Participants aged 18-49 years received placebo matched to RSV vaccine intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years: Participants aged 50-85 years received single 60-mcg dose of RSV vaccine, intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years: Participants aged 50-85 years received single 60-mcg dose with aluminum hydroxide intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 120 mcg Age 50-85 Years: Participants aged 50-85 years received single 120-mcg dose intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years: Participants aged 50-85 years received single 120-mcg dose with aluminum hydroxide intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 240 mcg Age 50-85 Years: Participants aged 50-85 years received single 240-mcg dose intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years: Participants aged 50-85 years received single 240-mcg dose with aluminum hydroxide intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: Placebo Age 50-85 Years: Participants aged 50-85 years received placebo matched to RSV vaccine intramuscularly. Participants were followed up to 12 months after vaccination.
- Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 60 mcg along with 0.5 milliliter (mL) seasonal inactivated influenza vaccine (SIIV) intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 60 mcg along with placebo (saline control) at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 60 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 60 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 120 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 120 mcg along with placebo (saline control) at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 120 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 120 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with placebo (saline control) at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV Intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV Intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received placebo (saline control) and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants who consented were revaccinated with placebo (saline control) and placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 60 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 60 mcg along with placebo (saline control) at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1.
- Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 60 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 60 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV Intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 120 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 120 mcg along with placebo (saline control) at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 120 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 120 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 240 mcg along with placebo (saline control) at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV Intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 240 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years: Participants aged 65-85 years received placebo (saline control) and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV intramuscularly at Day 35 (Vaccination 2). Participants who consented were revaccinated with placebo (saline control) and placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
Period: Overall Study
Arm/Group | Sentinel Cohort: Respiratory Syncytial Virus (RSV) Vaccine 60 Microgram (mcg) Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 41 | 42 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 40 | 42 | 40 | 40 | 41 | 41 | 40 | 41 | 42 | 43 | 41
Completed | 12 | 12 | 11 | 12 | 11 | 11 | 12 | 11 | 12 | 11 | 11 | 12 | 10 | 11 | 35 | 38 | 40 | 35 | 37 | 37 | 34 | 36 | 34 | 35 | 33 | 30 | 32 | 39 | 40 | 40 | 39 | 40 | 40 | 39 | 37 | 36 | 39 | 36 | 39 | 37
Not Completed | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 6 | 4 | 1 | 6 | 4 | 4 | 7 | 5 | 7 | 6 | 8 | 11 | 9 | 2 | 1 | 0 | 3 | 0 | 0 | 2 | 4 | 4 | 2 | 6 | 4 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 1 | 0 | 1 | 1 | 2 | 4 | 3 | 4 | 3 | 5 | 5 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 1
Not completed — No longer meets eligibility criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 3 | 1 | 3 | 1 | 1 | 2 | 2 | 4 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 1
Not completed — Screen Failure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Randomized but not vaccinated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants in the sentinel and expanded cohorts who received at least 1 dose of the investigational products.
Groups:
- Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years: Participants aged 18-49 years received single 60-mcg dose of RSV vaccine, intramuscularly. Participants were followed up to 12 months after vaccination.
- Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years; Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years: Participants aged 50-85 years received single 60-mcg dose with aluminum hydroxide intramuscularly. Participants were followed up to 12 months after vaccination.
- Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 60 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 120 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV Intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3) and received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Total: Total of all reporting groups
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 41 | 42 | 41 | 40 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 40 | 41 | 40 | 42 | 40 | 40 | 41 | 41 | 40 | 41 | 42 | 43 | 41 | 1233
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (9.5) | 34.0 (9.0) | 34.8 (8.0) | 34.2 (8.7) | 43.3 (4.8) | 36.3 (8.4) | 35.2 (9.4) | 65.4 (9.9) | 66.3 (9.7) | 63.7 (7.4) | 62.6 (8.6) | 62.1 (9.8) | 61.3 (7.7) | 61.3 (9.8) | 33.4 (8.2) | 32.6 (9.1) | 33.0 (8.6) | 34.1 (9.3) | 34.1 (8.5) | 36.8 (8.8) | 34.1 (8.7) | 33.1 (9.4) | 36.2 (8.9) | 34.7 (8.9) | 33.9 (8.5) | 34.6 (7.7) | 33.6 (8.5) | 72.6 (5.9) | 71.9 (4.8) | 72.4 (5.6) | 72.8 (5.1) | 70.9 (5.5) | 71.7 (5.4) | 72.2 (4.7) | 71.3 (4.8) | 72.3 (5.0) | 71.6 (5.2) | 71.4 (5.1) | 70.7 (4.9) | 70.9 (4.7) | 52.47 (19.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 6 | 10 | 9 | 9 | 5 | 7 | 8 | 7 | 5 | 10 | 9 | 6 | 27 | 28 | 27 | 25 | 29 | 29 | 26 | 25 | 29 | 29 | 28 | 29 | 29 | 17 | 23 | 20 | 25 | 24 | 22 | 22 | 23 | 26 | 26 | 26 | 20 | 29 | 771
  Male | 5 | 2 | 6 | 2 | 3 | 3 | 7 | 5 | 4 | 5 | 7 | 2 | 3 | 6 | 14 | 14 | 14 | 15 | 12 | 12 | 15 | 16 | 12 | 12 | 13 | 12 | 12 | 23 | 18 | 20 | 17 | 16 | 18 | 19 | 18 | 14 | 15 | 16 | 23 | 12 | 462
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 4 | 5 | 7 | 5 | 4 | 7 | 6 | 5 | 3 | 5 | 6 | 4 | 3 | 2 | 1 | 2 | 1 | 3 | 3 | 4 | 3 | 1 | 5 | 2 | 1 | 5 | 112
  Not Hispanic or Latino | 12 | 10 | 10 | 11 | 11 | 11 | 8 | 12 | 10 | 11 | 11 | 10 | 10 | 12 | 37 | 37 | 34 | 35 | 37 | 34 | 35 | 36 | 38 | 36 | 35 | 36 | 38 | 38 | 39 | 38 | 41 | 37 | 37 | 37 | 37 | 39 | 36 | 40 | 40 | 36 | 1112
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 10
  Asian | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Black or African American | 2 | 4 | 2 | 2 | 1 | 4 | 0 | 2 | 0 | 1 | 4 | 3 | 1 | 2 | 10 | 7 | 8 | 8 | 6 | 8 | 9 | 8 | 13 | 7 | 7 | 9 | 9 | 4 | 6 | 1 | 5 | 3 | 3 | 2 | 6 | 5 | 3 | 3 | 6 | 4 | 188
  White | 10 | 7 | 10 | 8 | 10 | 7 | 9 | 9 | 11 | 9 | 7 | 8 | 9 | 8 | 30 | 32 | 32 | 28 | 31 | 31 | 30 | 29 | 27 | 32 | 30 | 28 | 29 | 35 | 34 | 38 | 36 | 34 | 37 | 37 | 33 | 35 | 37 | 39 | 36 | 36 | 978
  More than one race | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 18 to 49 Years) With Local Reactions Within 14 Days After Vaccination
Description: Local reactions included pain at injection site, redness and swelling recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm) and graded as mild: 2.5 to 5.0 cm, moderate: greater than (>) 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfere with daily activity and severe: prevented daily activity.
Time Frame: Within 14 days after vaccination
Population: All participants in sentinel cohort who received at least 1 dose of the investigational products at Visit 1 and with e-dairy data available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 12 | 12
Percentage of participants
  Pain at injection site: mild | 50.0 [21.1 to 78.9] | 58.3 [27.7 to 84.8] | 25.0 [5.5 to 57.2] | 75.0 [42.8 to 94.5] | 0 [0.0 to 28.5] | 58.3 [27.7 to 84.8] | 16.7 [2.1 to 48.4]
  Pain at injection site: moderate | 0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 18.2 [2.3 to 51.8] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Pain at injection site: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Redness: mild | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Redness: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Redness: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Swelling: mild | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Swelling: moderate | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 28.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Swelling: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]

2. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 50 to 85 Years) With Local Reactions Within 14 Days After Vaccination
Description: Local reactions included pain at injection site, redness and swelling recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfered with daily activity and severe: prevented daily activity.
Time Frame: Within 14 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
Percentage of participants
  Pain at injection site: mild | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Pain at injection site: moderate | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 25.0 [5.5 to 57.2] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Pain at injection site: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Redness: mild | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Redness: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Redness: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Swelling: mild | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Swelling: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Swelling: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]

3. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 18 to 49 Years) With Local Reactions Within 14 Days After Vaccination 1
Description: Local reactions included pain at injection site, redness and swelling recorded by participants in an e-diary. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm and graded as mild: 2.5 to 5.0 cm, moderate: > 5.0 to 10.0 cm and severe: >10 cm. Pain at injection site was graded as mild: did not interfere with daily activity, moderate: interfere with daily activity and severe: prevented daily activity.
Time Frame: Within 14 days after vaccination 1 on Day 1
Population: All participants in expanded cohort who received at least 1 dose of the investigational products at Visit 1 and with e-dairy data available.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3). Participants received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with placebo (saline control) at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV Intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3). Participants received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3). Participants received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
- Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 240 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly at Day 1 (Vaccination 1). Participants received 0.5 mL SIIV Intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with aluminum hydroxide and placebo (saline control) intramuscularly after 12 months of Vaccination 1 (Vaccination 3). Participants received 0.5 mL SIIV intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 41 | 41 | 41 | 40 | 41 | 41 | 41 | 41 | 41
Percentage of participants
  Pain at injection site: mild | 34.1 [20.1 to 50.6] | 31.0 [17.6 to 47.1] | 41.5 [26.3 to 57.9] | 32.5 [18.6 to 49.1] | 36.6 [22.1 to 53.1] | 43.9 [28.5 to 60.3] | 48.8 [32.9 to 64.9] | 55.0 [38.5 to 70.7] | 24.4 [12.4 to 40.3] | 34.1 [20.1 to 50.6] | 51.2 [35.1 to 67.1] | 48.8 [32.9 to 64.9] | 14.6 [5.6 to 29.2]
  Pain at injection site: moderate | 12.2 [4.1 to 26.2] | 7.1 [1.5 to 19.5] | 26.8 [14.2 to 42.9] | 20.0 [9.1 to 35.6] | 9.8 [2.7 to 23.1] | 7.3 [1.5 to 19.9] | 12.2 [4.1 to 26.2] | 12.5 [4.2 to 26.8] | 14.6 [5.6 to 29.2] | 7.3 [1.5 to 19.9] | 9.8 [2.7 to 23.1] | 17.1 [7.2 to 32.1] | 2.4 [0.1 to 12.9]
  Pain at injection site: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6]
  Redness: mild | 2.4 [0.1 to 12.9] | 4.8 [0.6 to 16.2] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 7.5 [1.6 to 20.4] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 7.3 [1.5 to 19.9] | 4.9 [0.6 to 16.5] | 2.4 [0.1 to 12.9]
  Redness: moderate | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 4.9 [0.6 to 16.5] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 9.8 [2.7 to 23.1] | 0 [0.0 to 8.6]
  Redness: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6]
  Swelling: mild | 2.4 [0.1 to 12.9] | 4.8 [0.6 to 16.2] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 9.8 [2.7 to 23.1] | 2.4 [0.1 to 12.9] | 5.0 [0.6 to 16.9] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6] | 4.9 [0.6 to 16.5] | 9.8 [2.7 to 23.1] | 0 [0.0 to 8.6]
  Swelling: moderate | 2.4 [0.1 to 12.9] | 4.8 [0.6 to 16.2] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 7.3 [1.5 to 19.9] | 4.9 [0.6 to 16.5] | 2.4 [0.1 to 12.9] | 9.8 [2.7 to 23.1] | 0 [0.0 to 8.6]
  Swelling: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6]

4. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 65 to 85 Years) With Local Reactions Within 14 Days After Vaccination 1
Description: as for outcome 2
Time Frame: Within 14 days after vaccination 1 on Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years: Participants aged 65-85 years received RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1. Participants who consented were revaccinated with RSV vaccine 240 mcg along with 0.5 mL SIIV intramuscularly after 12 months of Vaccination 1 (Vaccination 3). Participants received placebo (saline control) intramuscularly at 35 days post Vaccination 3 (Vaccination 4). Participants were followed up to 12 months after Vaccination 3.
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Number analyzed (Participants) | 40 | 40 | 40 | 42 | 40 | 40 | 41 | 41 | 40 | 41 | 42 | 43 | 40
Percentage of participants
  Pain at injection site: mild | 25.0 [12.7 to 41.2] | 10.0 [2.8 to 23.7] | 22.5 [10.8 to 38.5] | 23.8 [12.1 to 39.5] | 22.5 [10.8 to 38.5] | 10.0 [2.8 to 23.7] | 26.8 [14.2 to 42.9] | 19.5 [8.8 to 34.9] | 32.5 [18.6 to 49.1] | 19.5 [8.8 to 34.9] | 19.0 [8.6 to 34.1] | 14.0 [5.3 to 27.9] | 5.0 [0.6 to 16.9]
  Pain at injection site: moderate | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 5.0 [0.6 to 16.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 4.8 [0.6 to 16.2] | 4.7 [0.6 to 15.8] | 0 [0.0 to 8.8]
  Pain at injection site: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Redness: mild | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 7.1 [1.5 to 19.5] | 2.5 [0.1 to 13.2] | 7.5 [1.6 to 20.4] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 7.3 [1.5 to 19.9] | 0 [0.0 to 8.4] | 4.7 [0.6 to 15.8] | 0 [0.0 to 8.8]
  Redness: moderate | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.6] | 5.0 [0.6 to 16.9] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.6] | 2.3 [0.1 to 12.3] | 0 [0.0 to 8.8]
  Redness: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Swelling: mild | 7.5 [1.6 to 20.4] | 5.0 [0.6 to 16.9] | 0 [0.0 to 8.8] | 4.8 [0.6 to 16.2] | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 5.0 [0.6 to 16.9] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.6] | 2.3 [0.1 to 12.3] | 2.5 [0.1 to 13.2]
  Swelling: moderate | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 5.0 [0.6 to 16.9] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.6] | 2.3 [0.1 to 12.3] | 0 [0.0 to 8.8]
  Swelling: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 2.3 [0.1 to 12.3] | 0 [0.0 to 8.8]

5. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 18 to 49 Years) With Systemic Reactions Within 14 Days After Vaccination
Description: Systemic reactions:fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever: greater than equal to (>=)38.0 degrees (deg) Celsius (C), mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 hours(h), moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
Time Frame: Within 14 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 12 | 12
Percentage of participants
  Fever: >=38.0 degree C | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Fever: mild | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fever: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Fever: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fever: Grade 4 | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fatigue: mild | 8.3 [0.2 to 38.5] | 41.7 [15.2 to 72.3] | 16.7 [2.1 to 48.4] | 33.3 [9.9 to 65.1] | 9.1 [0.2 to 41.3] | 16.7 [2.1 to 48.4] | 25.0 [5.5 to 57.2]
  Fatigue: moderate | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5] | 25.0 [5.5 to 57.2] | 25.0 [5.5 to 57.2] | 36.4 [10.9 to 69.2] | 33.3 [9.9 to 65.1] | 0 [0.0 to 26.5]
  Fatigue: severe | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 9.1 [0.2 to 41.3] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Headache: mild | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 33.3 [9.9 to 65.1] | 27.3 [6.0 to 61.0] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5]
  Headache: moderate | 25.0 [5.5 to 57.2] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 27.3 [6.0 to 61.0] | 33.3 [9.9 to 65.1] | 0 [0.0 to 26.5]
  Headache: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 9.1 [0.2 to 41.3] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Nausea: mild | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 28.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5]
  Nausea: moderate | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 18.2 [2.3 to 51.8] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Nausea: severe | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Muscle pain: mild | 50.0 [21.1 to 78.9] | 25.0 [5.5 to 57.2] | 25.0 [5.5 to 57.2] | 33.3 [9.9 to 65.1] | 0 [0.0 to 28.5] | 41.7 [15.2 to 72.3] | 8.3 [0.2 to 38.5]
  Muscle pain: moderate | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 9.1 [0.2 to 41.3] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5]
  Muscle pain: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 9.1 [0.2 to 41.3] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Joint pain: mild | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 28.5] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5]
  Joint pain: moderate | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 9.1 [0.2 to 41.3] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Joint pain: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 9.1 [0.2 to 41.3] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Vomiting: mild | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 18.2 [2.3 to 51.8] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Vomiting: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Vomiting: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Diarrhea: mild | 0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 27.3 [6.0 to 61.0] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Diarrhea: moderate | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5]
  Diarrhea: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 28.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]

6. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 50 to 85 Years) With Systemic Reactions Within 14 Days After Vaccination
Description: Systemic reactions: fever, fatigue/tiredness, headache, nausea, muscle pain, joint pain, vomiting, diarrhea and any systemic event recorded by participants in an e-diary. Fever: >= 38.0 deg C, mild (>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C), moderate (>38.9 to 40.0 deg C and >40.0 deg C), severe (>38.9 deg C to 40.0 deg C) and grade 4 (>40.0 deg C). Fatigue, headache, nausea, muscle pain and joint pain were graded as mild: did not interfere with activity, moderate: some interference with activity and severe: prevented daily routine activity. Vomiting was graded as mild: 1 to 2 times in 24 h, moderate: >2 times in 24h and severe: requires intravenous hydration. Diarrhea was graded as mild: 2 to 3 loose stools in 24h, moderate: 4 to 5 loose stools in 24h and severe: 6 or more loose stools in 24h.
Time Frame: Within 14 days after vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
Percentage of participants
  Fever: >=38.0 degree C | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fever: mild | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fever: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fever: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fever: Grade 4 | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Fatigue: mild | 41.7 [15.2 to 72.3] | 16.7 [2.1 to 48.4] | 33.3 [9.9 to 65.1] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4]
  Fatigue: moderate | 0 [0.0 to 26.5] | 33.3 [9.9 to 65.1] | 0 [0.0 to 26.5] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4]
  Fatigue: severe | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Headache: mild | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Headache: moderate | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5]
  Headache: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Nausea: mild | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Nausea: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Nausea: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Muscle pain: mild | 33.3 [9.9 to 65.1] | 33.3 [9.9 to 65.1] | 8.3 [0.2 to 38.5] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5] | 25.0 [5.5 to 57.2] | 0 [0.0 to 26.5]
  Muscle pain:moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5]
  Muscle pain: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Joint pain: mild | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Joint pain: moderate | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5]
  Joint pain: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Vomiting: mild | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Vomiting: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Vomiting: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]
  Diarrhea: mild | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5]
  Diarrhea: moderate | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5]
  Diarrhea: severe | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]

7. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 18 to 49 Years) With Systemic Reactions Within 14 Days After Vaccination 1
Description: as for outcome 6
Time Frame: Within 14 days after vaccination 1 on Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 41 | 41 | 41 | 40 | 41 | 41 | 41 | 41 | 41
Percentage of participants
  Fever: >=38.0 degree C | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 2.4 [0.1 to 12.9] | 2.5 [0.1 to 13.2] | 12.2 [4.1 to 26.2] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6]
  Fever: mild | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 4.9 [0.6 to 16.5] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6]
  Fever: moderate | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6]
  Fever: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6]
  Fever: Grade 4 | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6]
  Fatigue: mild | 14.6 [5.6 to 29.2] | 16.7 [7.0 to 31.4] | 17.1 [7.2 to 32.1] | 17.5 [7.3 to 32.8] | 17.1 [7.2 to 32.1] | 9.8 [2.7 to 23.1] | 29.3 [16.1 to 45.5] | 27.5 [14.6 to 43.9] | 14.6 [5.6 to 29.2] | 14.6 [5.6 to 29.2] | 29.3 [16.1 to 45.5] | 19.5 [8.8 to 34.9] | 12.2 [4.1 to 26.2]
  Fatigue: moderate | 31.7 [18.1 to 48.1] | 28.6 [15.7 to 44.6] | 24.4 [12.4 to 40.3] | 22.5 [10.8 to 38.5] | 19.5 [8.8 to 34.9] | 26.8 [14.2 to 42.9] | 14.6 [5.6 to 29.2] | 22.5 [10.8 to 38.5] | 29.3 [16.1 to 45.5] | 39.0 [24.2 to 55.5] | 19.5 [8.8 to 34.9] | 22.0 [10.6 to 37.6] | 19.5 [8.8 to 34.9]
  Fatigue: severe | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6]
  Headache: mild | 12.2 [4.1 to 26.2] | 28.6 [15.7 to 44.6] | 19.5 [8.8 to 34.9] | 32.5 [18.6 to 49.1] | 29.3 [16.1 to 45.5] | 17.1 [7.2 to 32.1] | 29.3 [16.1 to 45.5] | 27.5 [14.6 to 43.9] | 19.5 [8.8 to 34.9] | 7.3 [1.5 to 19.9] | 26.8 [14.2 to 42.9] | 24.4 [12.4 to 40.3] | 19.5 [8.8 to 34.9]
  Headache: moderate | 29.3 [16.1 to 45.5] | 21.4 [10.3 to 36.8] | 19.5 [8.8 to 34.9] | 10.0 [2.8 to 23.7] | 19.5 [8.8 to 34.9] | 24.4 [12.4 to 40.3] | 17.1 [7.2 to 32.1] | 20.0 [9.1 to 35.6] | 29.3 [16.1 to 45.5] | 29.3 [16.1 to 45.5] | 17.1 [7.2 to 32.1] | 14.6 [5.6 to 29.2] | 12.2 [4.1 to 26.2]
  Headache: severe | 2.4 [0.1 to 12.9] | 4.8 [0.6 to 16.2] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 7.3 [1.5 to 19.9] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6]
  Nausea: mild | 4.9 [0.6 to 16.5] | 7.1 [1.5 to 19.5] | 12.2 [4.1 to 26.2] | 12.5 [4.2 to 26.8] | 9.8 [2.7 to 23.1] | 19.5 [8.8 to 34.9] | 7.3 [1.5 to 19.9] | 7.5 [1.6 to 20.4] | 14.6 [5.6 to 29.2] | 14.6 [5.6 to 29.2] | 2.4 [0.1 to 12.9] | 9.8 [2.7 to 23.1] | 9.8 [2.7 to 23.1]
  Nausea: moderate | 9.8 [2.7 to 23.1] | 7.1 [1.5 to 19.5] | 7.3 [1.5 to 19.9] | 2.5 [0.1 to 13.2] | 4.9 [0.6 to 16.5] | 7.3 [1.5 to 19.9] | 4.9 [0.6 to 16.5] | 12.5 [4.2 to 26.8] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6] | 7.3 [1.5 to 19.9] | 7.3 [1.5 to 19.9] | 4.9 [0.6 to 16.5]
  Nausea: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6]
  Muscle pain: mild | 24.4 [12.4 to 40.3] | 16.7 [7.0 to 31.4] | 34.1 [20.1 to 50.6] | 27.5 [14.6 to 43.9] | 29.3 [16.1 to 45.5] | 22.0 [10.6 to 37.6] | 43.9 [28.5 to 60.3] | 37.5 [22.7 to 54.2] | 19.5 [8.8 to 34.9] | 24.4 [12.4 to 40.3] | 36.6 [22.1 to 53.1] | 26.8 [14.2 to 42.9] | 12.2 [4.1 to 26.2]
  Muscle pain: moderate | 14.6 [5.6 to 29.2] | 14.3 [5.4 to 28.5] | 22.0 [10.6 to 37.6] | 10.0 [2.8 to 23.7] | 4.9 [0.6 to 16.5] | 19.5 [8.8 to 34.9] | 17.1 [7.2 to 32.1] | 12.5 [4.2 to 26.8] | 19.5 [8.8 to 34.9] | 12.2 [4.1 to 26.2] | 7.3 [1.5 to 19.9] | 19.5 [8.8 to 34.9] | 0 [0.0 to 8.6]
  Muscle pain: severe | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 4.9 [0.6 to 16.5] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6]
  Joint pain: mild | 12.2 [4.1 to 26.2] | 4.8 [0.6 to 16.2] | 14.6 [5.6 to 29.2] | 2.5 [0.1 to 13.2] | 12.2 [4.1 to 26.2] | 4.9 [0.6 to 16.5] | 14.6 [5.6 to 29.2] | 12.5 [4.2 to 26.8] | 7.3 [1.5 to 19.9] | 4.9 [0.6 to 16.5] | 9.8 [2.7 to 23.1] | 7.3 [1.5 to 19.9] | 4.9 [0.6 to 16.5]
  Joint pain: moderate | 7.3 [1.5 to 19.9] | 7.1 [1.5 to 19.5] | 9.8 [2.7 to 23.1] | 2.5 [0.1 to 13.2] | 7.3 [1.5 to 19.9] | 7.3 [1.5 to 19.9] | 9.8 [2.7 to 23.1] | 17.5 [7.3 to 32.8] | 9.8 [2.7 to 23.1] | 12.2 [4.1 to 26.2] | 7.3 [1.5 to 19.9] | 9.8 [2.7 to 23.1] | 0 [0.0 to 8.6]
  Joint pain: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6]
  Vomiting: mild | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9]
  Vomiting: moderate | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6]
  Vomiting: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6]
  Diarrhea: mild | 7.3 [1.5 to 19.9] | 11.9 [4.0 to 25.6] | 19.5 [8.8 to 34.9] | 12.5 [4.2 to 26.8] | 22.0 [10.6 to 37.6] | 17.1 [7.2 to 32.1] | 19.5 [8.8 to 34.9] | 22.5 [10.8 to 38.5] | 12.2 [4.1 to 26.2] | 19.5 [8.8 to 34.9] | 7.3 [1.5 to 19.9] | 17.1 [7.2 to 32.1] | 9.8 [2.7 to 23.1]
  Diarrhea: moderate | 7.3 [1.5 to 19.9] | 11.9 [4.0 to 25.6] | 4.9 [0.6 to 16.5] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 7.3 [1.5 to 19.9] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 4.9 [0.6 to 16.5] | 7.3 [1.5 to 19.9] | 2.4 [0.1 to 12.9]
  Diarrhea: severe | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6]

8. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 65 to 85 Years) With Systemic Reactions Within 14 Days After Vaccination 1
Description: as for outcome 6
Time Frame: Within 14 days after vaccination 1 on Day 1
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Number analyzed (Participants) | 40 | 40 | 40 | 42 | 40 | 40 | 41 | 41 | 40 | 41 | 42 | 43 | 40
Percentage of participants
  Fever: >=38.0 degree C | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 4.8 [0.6 to 16.2] | 4.7 [0.6 to 15.8] | 0 [0.0 to 8.8]
  Fever: mild | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 4.8 [0.6 to 16.2] | 2.3 [0.1 to 12.3] | 0 [0.0 to 8.8]
  Fever: moderate | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 2.3 [0.1 to 12.3] | 0 [0.0 to 8.8]
  Fever: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Fever: Grade 4 | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Fatigue: mild | 7.5 [1.6 to 20.4] | 12.5 [4.2 to 26.8] | 12.5 [4.2 to 26.8] | 26.2 [13.9 to 42.0] | 10.0 [2.8 to 23.7] | 7.5 [1.6 to 20.4] | 14.6 [5.6 to 29.2] | 14.6 [5.6 to 29.2] | 22.5 [10.8 to 38.5] | 19.5 [8.8 to 34.9] | 23.8 [12.1 to 39.5] | 20.9 [10.0 to 36.0] | 7.5 [1.6 to 20.4]
  Fatigue: moderate | 12.5 [4.2 to 26.8] | 10.0 [2.8 to 23.7] | 15.0 [5.7 to 29.8] | 11.9 [4.0 to 25.6] | 12.5 [4.2 to 26.8] | 10.0 [2.8 to 23.7] | 19.5 [8.8 to 34.9] | 14.6 [5.6 to 29.2] | 20.0 [9.1 to 35.6] | 4.9 [0.6 to 16.5] | 21.4 [10.3 to 36.8] | 4.7 [0.6 to 15.8] | 7.5 [1.6 to 20.4]
  Fatigue: severe | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.6] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Headache: mild | 17.5 [7.3 to 32.8] | 7.5 [1.6 to 20.4] | 7.5 [1.6 to 20.4] | 14.3 [5.4 to 28.5] | 15.0 [5.7 to 29.8] | 12.5 [4.2 to 26.8] | 7.3 [1.5 to 19.9] | 22.0 [10.6 to 37.6] | 10.0 [2.8 to 23.7] | 24.4 [12.4 to 40.3] | 21.4 [10.3 to 36.8] | 9.3 [2.6 to 22.1] | 20.0 [9.1 to 35.6]
  Headache: moderate | 7.5 [1.6 to 20.4] | 5.0 [0.6 to 16.9] | 5.0 [0.6 to 16.9] | 2.4 [0.1 to 12.6] | 2.5 [0.1 to 13.2] | 5.0 [0.6 to 16.9] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 5.0 [0.6 to 16.9] | 2.4 [0.1 to 12.9] | 11.9 [4.0 to 25.6] | 11.6 [3.9 to 25.1] | 2.5 [0.1 to 13.2]
  Headache: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Nausea: mild | 5.0 [0.6 to 16.9] | 7.5 [1.6 to 20.4] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.4] | 5.0 [0.6 to 16.9] | 5.0 [0.6 to 16.9] | 7.3 [1.5 to 19.9] | 4.9 [0.6 to 16.5] | 7.5 [1.6 to 20.4] | 9.8 [2.7 to 23.1] | 2.4 [0.1 to 12.6] | 2.3 [0.1 to 12.3] | 5.0 [0.6 to 16.9]
  Nausea: moderate | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 14.6 [5.6 to 29.2] | 5.0 [0.6 to 16.9] | 0 [0.0 to 8.6] | 4.8 [0.6 to 16.2] | 2.3 [0.1 to 12.3] | 0 [0.0 to 8.8]
  Nausea: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Muscle pain: mild | 15.0 [5.7 to 29.8] | 7.5 [1.6 to 20.4] | 10.0 [2.8 to 23.7] | 14.3 [5.4 to 28.5] | 15.0 [5.7 to 29.8] | 5.0 [0.6 to 16.9] | 14.6 [5.6 to 29.2] | 19.5 [8.8 to 34.9] | 17.5 [7.3 to 32.8] | 17.1 [7.2 to 32.1] | 19.0 [8.6 to 34.1] | 4.7 [0.6 to 15.8] | 7.5 [1.6 to 20.4]
  Muscle pain: moderate | 2.5 [0.1 to 13.2] | 7.5 [1.6 to 20.4] | 5.0 [0.6 to 16.9] | 2.4 [0.1 to 12.6] | 7.5 [1.6 to 20.4] | 7.5 [1.6 to 20.4] | 4.9 [0.6 to 16.5] | 4.9 [0.6 to 16.5] | 15.0 [5.7 to 29.8] | 9.8 [2.7 to 23.1] | 16.7 [7.0 to 31.4] | 16.3 [6.8 to 30.7] | 0 [0.0 to 8.8]
  Muscle pain: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 2.5 [0.1 to 13.2]
  Joint pain: mild | 12.5 [4.2 to 26.8] | 10.0 [2.8 to 23.7] | 5.0 [0.6 to 16.9] | 9.5 [2.7 to 22.6] | 10.0 [2.8 to 23.7] | 7.5 [1.6 to 20.4] | 7.3 [1.5 to 19.9] | 7.3 [1.5 to 19.9] | 12.5 [4.2 to 26.8] | 7.3 [1.5 to 19.9] | 21.4 [10.3 to 36.8] | 2.3 [0.1 to 12.3] | 7.5 [1.6 to 20.4]
  Joint pain: moderate | 7.5 [1.6 to 20.4] | 5.0 [0.6 to 16.9] | 5.0 [0.6 to 16.9] | 9.5 [2.7 to 22.6] | 5.0 [0.6 to 16.9] | 7.5 [1.6 to 20.4] | 4.9 [0.6 to 16.5] | 7.3 [1.5 to 19.9] | 0 [0.0 to 8.8] | 9.8 [2.7 to 23.1] | 7.1 [1.5 to 19.5] | 4.7 [0.6 to 15.8] | 7.5 [1.6 to 20.4]
  Joint pain: severe | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Vomiting: mild | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 2.4 [0.1 to 12.9] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 2.3 [0.1 to 12.3] | 0 [0.0 to 8.8]
  Vomiting: moderate | 0 [0.0 to 8.8] | 2.5 [0.1 to 13.2] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 4.9 [0.6 to 16.5] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Vomiting: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.4] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.2] | 0 [0.0 to 8.8]
  Diarrhea: mild | 5.0 [0.6 to 16.9] | 15.0 [5.7 to 29.8] | 20.0 [9.1 to 35.6] | 7.1 [1.5 to 19.5] | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 7.3 [1.5 to 19.9] | 7.3 [1.5 to 19.9] | 17.5 [7.3 to 32.8] | 7.3 [1.5 to 19.9] | 14.3 [5.4 to 28.5] | 2.3 [0.1 to 12.3] | 5.0 [0.6 to 16.9]
  Diarrhea: moderate | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.6] | 5.0 [0.6 to 16.9] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 7.3 [1.5 to 19.9] | 7.5 [1.6 to 20.4] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 4.7 [0.6 to 15.8] | 0 [0.0 to 8.8]
  Diarrhea: severe | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.6] | 0 [0.0 to 8.8] | 0 [0.0 to 8.8] | 0 [0.0 to 8.6] | 0 [0.0 to 8.6] | 0 [0.0 to 8.8] | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 2.3 [0.1 to 12.3] | 2.5 [0.1 to 13.2]

9. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 18 to 49 Years) With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Within 1 month after vaccination (up to 35 days)
Population: All participants in sentinel cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
Percentage of participants | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5]

10. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 50 to 85 Years) With AEs Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Within 1 month after vaccination (up to 35 days)
Population: All participants in sentinel cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
Percentage of participants | 25.0 [5.5 to 57.2] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]

11. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 18 to 49 Years) With AE Within 1 Month After Vaccination 1
Description: as for outcome 10
Time Frame: Within 1 month after vaccination 1 (up to 35 days)
Population: All participants in expanded cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41
Percentage of participants | 17.1 [7.2 to 32.1] | 16.7 [7.0 to 31.4] | 14.6 [5.6 to 29.2] | 22.5 [10.8 to 38.5] | 24.4 [12.4 to 40.3] | 22.0 [10.6 to 37.6] | 7.3 [1.5 to 19.9] | 22.0 [10.6 to 37.6] | 9.8 [2.7 to 23.1] | 12.2 [4.1 to 26.2] | 12.2 [4.1 to 26.2] | 17.1 [7.2 to 32.1] | 9.8 [2.7 to 23.1]

12. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 65 to 85 Years) With AE Within 1 Month After Vaccination
Description: as for outcome 10
Time Frame: Within 1 month after vaccination 1 (up to 35 days)
Population: All participants in expanded cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Number analyzed (Participants) | 40 | 41 | 40 | 42 | 40 | 40 | 41 | 41 | 40 | 41 | 42 | 43 | 41
Percentage of participants | 10.0 [2.8 to 23.7] | 14.6 [5.6 to 29.2] | 5.0 [0.6 to 16.9] | 26.2 [13.9 to 42.0] | 22.5 [10.8 to 38.5] | 20.0 [9.1 to 35.6] | 14.6 [5.6 to 29.2] | 14.6 [5.6 to 29.2] | 15.0 [5.7 to 29.8] | 9.8 [2.7 to 23.1] | 11.9 [4.0 to 25.6] | 16.3 [6.8 to 30.7] | 12.2 [4.1 to 26.2]

13. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 18 to 49 Years) With Medically Attended Adverse Events (MAEs) and Serious Adverse Events (SAEs) Upto 12 Months After Vaccination
Description: MAE was defined as a non-serious AE that resulted in an evaluation at a medical facility. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Upto 12 months after vaccination (up to 378 days)
Population: All participants in sentinel cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
Percentage of participants
  MAEs | 33.3 [9.9 to 65.1] | 0 [0.0 to 26.5] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4]
  SAEs | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5]

14. Primary Outcome: Sentinel Cohort: Percentage of Participants (Aged 50 to 85 Years) With MAEs and SAEs Upto 12 Months After Vaccination
Description: as for outcome 13
Time Frame: Upto 12 months after vaccination (upto 378 days)
Population: All participants in sentinel cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years:: Participants aged 50-85 years received single 60-mcg dose of RSV vaccine, intramuscularly. Participants were followed up to 12 months after vaccination.
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years: | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12
Percentage of participants
  MAEs | 25.0 [5.5 to 57.2] | 50.0 [21.1 to 78.9] | 25.0 [5.5 to 57.2] | 25.0 [5.5 to 57.2] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4]
  SAEs | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 0 [0.0 to 26.5] | 8.3 [0.2 to 38.5] | 16.7 [2.1 to 48.4] | 0 [0.0 to 26.5]

15. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 18 to 49 Years) With MAEs and SAEs Upto 12 Months After Vaccination 1
Description: as for outcome 13
Time Frame: Upto 12 months after vaccination 1 (upto 378 days)
Population: All participants in expanded cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41
Percentage of participants
  MAEs | 22.0 [10.6 to 37.6] | 14.3 [5.4 to 28.5] | 9.8 [2.7 to 23.1] | 17.5 [7.3 to 32.8] | 22.0 [10.6 to 37.6] | 19.5 [8.8 to 34.9] | 12.2 [4.1 to 26.2] | 24.4 [12.4 to 40.3] | 24.4 [12.4 to 40.3] | 22.0 [10.6 to 40.3] | 24.4 [12.4 to 40.3] | 22.0 [10.6 to 37.6] | 22.0 [10.6 to 37.6]
  SAEs | 2.4 [0.1 to 12.9] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6] | 2.5 [0.1 to 13.2] | 2.4 [0.1 to 12.9] | 4.9 [0.6 to 16.5] | 0 [0.0 to 8.6] | 4.9 [0.6 to 16.5] | 4.9 [0.6 to 16.5] | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.9] | 7.3 [1.5 to 19.9] | 2.4 [0.1 to 12.9]

16. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 65 to 85 Years) With MAEs and SAEs 12 Months After Vaccination 1
Description: as for outcome 13
Time Frame: Upto 12 months after vaccination 1 (upto 378 days)
Population: All participants in expanded cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Number analyzed (Participants) | 40 | 41 | 40 | 42 | 40 | 40 | 41 | 41 | 40 | 41 | 42 | 43 | 41
Percentage of participants
  MAEs | 15.0 [5.7 to 29.8] | 24.4 [12.4 to 40.3] | 30.0 [16.6 to 46.5] | 31.0 [17.6 to 47.1] | 22.5 [10.8 to 38.5] | 22.5 [10.8 to 38.5] | 17.1 [7.2 to 32.1] | 34.1 [20.1 to 50.6] | 47.5 [31.5 to 63.9] | 43.9 [28.5 to 60.3] | 28.6 [15.7 to 44.6] | 25.6 [13.5 to 41.2] | 14.6 [5.6 to 29.2]
  SAEs | 5.0 [0.6 to 16.9] | 17.1 [7.2 to 32.1] | 10.0 [2.8 to 23.7] | 19.0 [8.6 to 34.1] | 10.0 [2.8 to 23.7] | 5.0 [0.6 to 16.9] | 17.1 [7.2 to 32.1] | 4.9 [0.6 to 16.5] | 10.0 [2.8 to 23.7] | 7.3 [1.5 to 19.9] | 7.1 [1.5 to 19.5] | 7.0 [1.5 to 19.1] | 7.3 [1.5 to 19.9]

17. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 18 to 49 Years) With AEs Within 1 Month After Vaccination 2
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events.
Time Frame: Within 1 month after vaccination 2 (upto Day 70)
Population: All participants in expanded cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years
Number analyzed (Participants) | 41 | 42 | 41 | 40 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41 | 41
Percentage of participants | 19.5 [8.8 to 34.9] | 14.3 [5.4 to 28.5] | 19.5 [8.8 to 34.9] | 10.0 [2.8 to 23.7] | 7.3 [1.5 to 19.9] | 17.1 [7.2 to 32.1] | 22.0 [10.6 to 37.6] | 14.6 [5.6 to 29.2] | 26.8 [14.2 to 42.9] | 26.8 [14.2 to 42.9] | 19.5 [8.8 to 34.9] | 17.1 [7.2 to 32.1] | 9.8 [2.7 to 23.1]

18. Primary Outcome: Expanded Cohort: Percentage of Participants (Aged 65 to 85 Years) With AEs Within 1 Month After Vaccination 2
Description: as for outcome 17
Time Frame: Within 1 month after vaccination 2 (upto Day 70)
Population: All participants in expanded cohort who received at least 1 dose of the investigational products at Visit 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Number analyzed (Participants) | 40 | 41 | 40 | 42 | 40 | 40 | 41 | 41 | 40 | 41 | 42 | 43 | 41
Percentage of participants | 10.0 [2.8 to 23.7] | 7.3 [1.5 to 19.9] | 20.0 [9.1 to 35.6] | 21.4 [10.3 to 36.8] | 25.0 [12.7 to 41.2] | 30.0 [16.6 to 46.5] | 12.2 [4.1 to 26.2] | 9.8 [2.7 to 23.1] | 32.5 [18.6 to 49.1] | 24.4 [12.4 to 40.3] | 11.9 [4.0 to 25.6] | 18.6 [8.4 to 33.4] | 17.1 [7.2 to 32.1]

19. Secondary Outcome: Sentinel Cohort: Geometric Mean Titers (GMTs) of Respiratory Syncytial Virus Subgroup A (RSV A) and RSV B Antigens Following Vaccination in Participants (Aged 18 to 49 Years)
Description: GMTs of RSV A and RSV B antigens were measured using neutralizing assay. The neutralizing titer lower limit of quantitation (LLOQ) values were: A = 50 and B = 70. Assay results below the LLOQ were set to 0.5*LLOQ. Titers were expressed in terms of 1/dilution.
Time Frame: Before vaccination, and 2 weeks and 1, 2, 3, 6 and 12 months after vaccination
Population: Evaluable immunogenicity population (EIP): participants who were eligible, received all RSV vaccine or placebo to which they were randomized, had blood drawn for assay testing within 27 to 42 days after Visit 1, had at least 1 valid and determinate assay result at 1-month-postvaccination visit and no major protocol violations. Here, "number analyzed" signifies participants evaluable at specific rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 11 | 11 | 12
Titers
  RSV A: before vaccination 1 | 1319 [639.4 to 2720.0] | 1754 [1053.6 to 2919.0] | 1090 [636.6 to 1867.2] | 1531 [939.0 to 2495.5] | 2029 [1186.2 to 3471.1] | 1553 [997.5 to 2416.8] | 1229 [666.0 to 2267.8]
  RSV A: 2 Weeks after vaccination 1 | 20936 [16760.8 to 26151.7] | 24970 [15120.8 to 41235.7] | 31584 [19599.9 to 50897.0] | 31193 [18221.6 to 53399.1] | 44866 [27431.6 to 73379.3] | 52339 [41244.0 to 66419.5] | 2817 [1279.8 to 6200.0]
  RSV A: 1 Month after vaccination 1 | 16730 [10482.1 to 26701.2] | 20512 [10692.1 to 39349.2] | 10021 [5439.7 to 18461.5] | 16521 [8363.4 to 32634.1] | 27892 [11836.8 to 65726.0] | 28453 [17960.2 to 45076.0] | 2430 [1059.5 to 5572.8]
  RSV A: 2 Months after vaccination 1 | 12702 [7774.1 to 20752.2] | 28577 [17569.4 to 46482.7] | 11171 [7299.6 to 17095.6] | 15529 [8421.5 to 28636.3] | 23033 [15199.1 to 34905.6] | 18883 [11903.1 to 29955.5] | 1851 [872.8 to 3925.5]
  RSV A:3 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 11 | 12 | 11 | 11 | 12
  RSV A:3 Months after vaccination 1 | 8258 [5436.7 to 12544.3] | 15276 [8311.3 to 28077.4] | 10800 [5629.4 to 20720.5] | 12421 [6536.5 to 23602.4] | 19654 [11887.0 to 32494.6] | 12922 [8416.3 to 19839.5] | 1560 [871.7 to 2791.5]
  RSV A:6 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 10 | 12 | 11 | 11 | 12
  RSV A:6 Months after vaccination 1 | 11466 [7413.8 to 17733.3] | 22737 [13621.9 to 37952.6] | 12034 [6531.3 to 22173.9] | 9707 [5968.0 to 15788.1] | 13672 [8854.3 to 21111.5] | 8237 [5457.7 to 12430.7] | 2658 [1713.6 to 4121.5]
  RSV A: 12 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 11 | 12 | 11 | 11 | 12
  RSV A: 12 Months after vaccination 1 | 4430 [1406.2 to 13954.0] | 11052 [6489.0 to 18822.7] | 6147 [3027.2 to 12480.5] | 5849 [2465.2 to 13876.7] | 9851 [6172.1 to 15722.6] | 8707 [5584.9 to 13573.9] | 2043 [1043.0 to 4002.1]
  RSV B: before vaccination 1 | 1427 [696.9 to 2921.5] | 2077 [1318.2 to 3274.2] | 995 [468.6 to 2111.4] | 1670 [987.2 to 2826.2] | 1600 [884.5 to 2895.1] | 1492 [946.5 to 2353.0] | 1393 [600.9 to 3227.2]
  RSV B: 2 Weeks after vaccination 1 | 23974 [17227.4 to 33364.1] | 22491 [12970.4 to 38999.0] | 32104 [22689.9 to 45424.2] | 42222 [18956.4 to 94043.4] | 59752 [32986.4 to 108235.8] | 59955 [39010.7 to 92143.8] | 2817 [1109.7 to 7150.1]
  RSV B: 1 Month after vaccination 1 | 18932 [11958.2 to 29973.5] | 19197 [9637.0 to 38241.0] | 8510 [5282.6 to 13708.4] | 18080 [8223.8 to 39749.5] | 26759 [10616.0 to 67451.3] | 29668 [17559.4 to 50125.0] | 1861 [657.4 to 5265.8]
  RSV B: 2 Months after vaccination 1 | 13959 [8783.3 to 22184.4] | 28374 [15306.1 to 52600.1] | 8760 [5253.7 to 14607.8] | 16167 [7902.3 to 33077.1] | 19534 [10586.7 to 36042.0] | 18280 [10621.2 to 31462.6] | 1604 [606.9 to 4238.4]
  RSV B: 3 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 11 | 12 | 11 | 11 | 12
  RSV B: 3 Months after vaccination 1 | 9688 [6307.1 to 14882.3] | 12697 [7257.0 to 22214.4] | 8833 [5170.6 to 15088.1] | 11986 [5852.2 to 24549.6] | 16706 [8822.8 to 31633.4] | 11588 [6572.0 to 20434.1] | 1613 [780.6 to 3331.5]
  RSV B: 6 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 10 | 12 | 11 | 11 | 12
  RSV B: 6 Months after vaccination 1 | 15235 [7604.2 to 30523.5] | 16492 [10319.2 to 26357.8] | 10918 [5615.7 to 21225.9] | 11658 [6759.2 to 20107.4] | 11857 [6383.5 to 22021.8] | 7435 [4660.4 to 11862.2] | 2865 [1655.5 to 4960.0]
  RSV B: 12 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 11 | 12 | 11 | 11 | 12
  RSV B: 12 Months after vaccination 1 | 4674 [1561.6 to 13991.5] | 9274 [5661.4 to 15192.8] | 4127 [2331.4 to 7303.9] | 5392 [2058.4 to 14125.8] | 8565 [4633.3 to 15832.7] | 7373 [4569.2 to 11897.9] | 1970 [839.1 to 4625.6]

20. Secondary Outcome: Sentinel Cohort: GMTs of RSV A and RSV B Antigens Following Vaccination in Participants (Aged 50 to 85 Years)
Description: GMTs of RSV A and RSV B antigens were measured using neutralizing assay. The neutralizing titer LLOQ values were: A = 50 and B = 70. Assay results below the LLOQ were set to 0.5*LLOQ. Titers were expressed in terms of 1/dilution.
Time Frame: Before vaccination, and 2 weeks and 1, 2, 3, 6 and 12 months after vaccination
Population: EIP: participants who were eligible, received all RSV vaccine or placebo to which they were randomized, had blood drawn for assay testing within 27 to 42 days after Visit 1, had at least 1 valid and determinate assay result at 1-month-postvaccination visit and no major protocol violations. Here, "number analyzed" signifies participants evaluable at specific rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 11
Titers
  RSV A: before vaccination 1 | 1904 [1278.7 to 2834.4] | 1672 [1040.7 to 2686.7] | 2056 [1331.2 to 3173.9] | 1923 [1005.6 to 3678.3] | 1923 [1336.2 to 2766.2] | 1564 [937.6 to 2607.5] | 2359 [1410.7 to 3943.4]
  RSV A: 2 Weeks after vaccination 1 | 17464 [8895.2 to 34285.4] | 22594 [11704.0 to 43617.7] | 31946 [20617.5 to 49500.7] | 30618 [19555.9 to 47936.7] | 29812 [19802.0 to 44882.0] | 40272 [21945.3 to 73902.5] | 2233 [1688.2 to 2953.0]
  RSV A: 1 Month after vaccination 1 | 21116 [10249.1 to 43505.0] | 21788 [13645.3 to 34789.6] | 23161 [13893.6 to 38609.1] | 20499 [14652.3 to 28677.5] | 24481 [14704.5 to 40757.9] | 36197 [23048.4 to 56845.6] | 2675 [1318.3 to 5428.2]
  RSV A: 2 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 12 | 11
  RSV A: 2 Months after vaccination 1 | 15025 [7591.1 to 29738.7] | 10949 [6413.2 to 18694.3] | 16441 [10140.5 to 26656.3] | 10493 [6930.9 to 15884.4] | 12659 [8728.3 to 18358.5] | 13723 [6897.6 to 27300.9] | 1502 [1051.7 to 2143.7]
  RSV A:3 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 11 | 11
  RSV A:3 Months after vaccination 1 | 9792 [5705.9 to 16804.9] | 12202 [8157.6 to 18250.8] | 11476 [6917.1 to 19038.6] | 11561 [6851.2 to 19508.3] | 11195 [7550.0 to 16599.6] | 12747 [5865.4 to 27701.7] | 1543 [1045.0 to 2276.9]
  RSV A:6 Months after vaccination 1: number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 11 | 11
  RSV A:6 Months after vaccination 1 | 12290 [6656.1 to 22693.9] | 10213 [6473.8 to 16111.2] | 12795 [8778.0 to 18649.5] | 12172 [6876.4 to 21545.6] | 7083 [4674.4 to 10732.7] | 9417 [5251.7 to 16885.6] | 1945 [1081.1 to 3498.6]
  RSV A: 12 Months after vaccination 1: number analyzed (Participants) | 11 | 12 | 11 | 11 | 12 | 10 | 10
  RSV A: 12 Months after vaccination 1 | 9446 [5677.6 to 15715.0] | 7507 [4093.7 to 13766.5] | 8484 [5809.9 to 12390.3] | 10709 [6444.0 to 17798.1] | 2705 [644.6 to 11353.2] | 4145 [1867.0 to 9204.4] | 2341 [1216.8 to 4502.5]
  RSV B: before vaccination 1 | 2573 [1589.0 to 4166.1] | 1139 [693.5 to 1871.0] | 1190 [670.8 to 2111.9] | 1568 [755.8 to 3254.9] | 2144 [1317.6 to 3490.2] | 1417 [872.5 to 2301.3] | 2285 [1440.4 to 3624.1]
  RSV B: 2 Weeks after vaccination 1 | 27923 [14883.3 to 52385.8] | 19751 [10180.1 to 38319.0] | 25820 [11849.7 to 56262.2] | 33779 [19683.4 to 57969.0] | 47514 [26993.7 to 83633.1] | 41776 [20962.6 to 83256.1] | 2441 [1741.5 to 3421.0]
  RSV B: 1 Month after vaccination 1 | 27789 [14463.8 to 53392.0] | 21429 [10960.1 to 41899.2] | 16610 [7522.2 to 36678.1] | 19632 [13014.2 to 29615.5] | 32668 [18110.7 to 58926.6] | 37852 [22637.3 to 63291.6] | 3104 [1630.2 to 5908.9]
  RSV B: 2 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 12 | 11
  RSV B: 2 Months after vaccination 1 | 19061 [9784.0 to 37133.0] | 10713 [5704.5 to 20118.3] | 11284 [5285.1 to 24091.8] | 9247 [5754.6 to 14860.4] | 15567 [9281.5 to 26110.1] | 12441 [7391.4 to 20941.9] | 1461 [995.6 to 2143.4]
  RSV B: 3 Months after vaccination 1: number analyzed (Participants) | 12 | 12 | 12 | 11 | 12 | 11 | 11
  RSV B: 3 Months after vaccination 1 | 12225 [5963.9 to 25058.3] | 10364 [5186.7 to 20708.8] | 7190 [3217.8 to 16066.1] | 11138 [6751.8 to 18373.7] | 12998 [7277.3 to 23215.1] | 11726 [6130.9 to 22427.1] | 1436 [938.4 to 2196.9]
  RSV B: 6 Months after vaccination 1: number analyzed (Participants) | 11 | 12 | 12 | 11 | 12 | 11 | 11
  RSV B: 6 Months after vaccination 1 | 16998 [7585.9 to 38087.5] | 11281 [6198.0 to 20531.5] | 8636 [4397.3 to 16960.1] | 12541 [6303.2 to 24951.9] | 6949 [4175.8 to 11565.2] | 8066 [4681.5 to 13896.6] | 1920 [1307.0 to 2821.0]
  RSV B: 12 Months after vaccination 1: number analyzed (Participants) | 11 | 12 | 11 | 11 | 12 | 10 | 10
  RSV B: 12 Months after vaccination 1 | 9721 [4894.4 to 19308.4] | 5801 [3688.7 to 9122.8] | 6174 [3406.1 to 11192.6] | 8589 [4898.5 to 15059.1] | 3230 [765.7 to 13626.8] | 2918 [855.6 to 9948.1] | 2188 [1398.7 to 3423.8]

21. Secondary Outcome: Expanded Cohort: GMTs of RSV A and RSV B Antigens Following Vaccination in Participants (Aged 18 to 49 Years)
Description: as for outcome 20
Time Frame: Before vaccination, 1, 2, 3, 6 and 12 months after vaccination
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years
Number analyzed (Participants) | 39 | 39 | 40 | 38 | 40 | 40 | 39 | 38 | 40 | 39 | 41 | 40 | 41
Titers
  RSV A: before vaccination 1 | 1998 [1544.9 to 2583.6] | 1471 [1136.8 to 1904.1] | 1518 [1124.2 to 2049.1] | 1768 [1355.5 to 2305.0] | 1297 [995.4 to 1689.3] | 1713 [1288.9 to 2276.8] | 1862 [1443.5 to 2402.8] | 1933 [1531.1 to 2440.5] | 1733 [1352.7 to 2220.3] | 1640 [1175.5 to 2289.3] | 1522 [1162.6 to 1991.9] | 1625 [1209.9 to 2183.4] | 1750 [1398.4 to 2190.0]
  RSV A: 1 Month after vaccination 1 | 17482 [13630.9 to 22420.4] | 21728 [17712.2 to 26655.0] | 17460 [12975.9 to 23494.5] | 18064 [13868.8 to 23527.5] | 17760 [13990.9 to 22544.3] | 22628 [17718.2 to 28899.1] | 26465 [20604.2 to 33993.1] | 25860 [18817.4 to 35539.3] | 23783 [18268.5 to 30962.6] | 29332 [24173.0 to 35591.1] | 21196 [15702.1 to 28611.6] | 26938 [20516.3 to 35369.1] | 1883 [1465.0 to 2419.5]
  RSV A: 2 Months after vaccination 1: number analyzed (Participants) | 38 | 38 | 39 | 38 | 39 | 39 | 39 | 35 | 40 | 39 | 39 | 38 | 41
  RSV A: 2 Months after vaccination 1 | 10247 [8239.7 to 12743.8] | 11976 [9521.6 to 15064.2] | 10326 [7936.9 to 13433.2] | 12522 [9469.3 to 16557.6] | 9595 [7224.8 to 12743.7] | 14140 [11050.3 to 18093.4] | 15754 [11605.8 to 21383.9] | 13518 [10423.6 to 17530.1] | 13790 [10401.4 to 18281.4] | 14999 [11660.3 to 19294.4] | 11533 [8867.3 to 14999.7] | 12812 [9507.1 to 17265.5] | 1252 [988.9 to 1584.0]
  RSV A:3 Months after vaccination 1: number analyzed (Participants) | 37 | 38 | 39 | 38 | 38 | 38 | 39 | 35 | 40 | 39 | 40 | 38 | 41
  RSV A:3 Months after vaccination 1 | 11164 [8453.8 to 14743.3] | 12664 [10280.1 to 15600.9] | 12042 [9262.7 to 15655.6] | 12773 [9651.2 to 16903.6] | 9205 [7081.5 to 11965.6] | 13801 [10058.5 to 18934.9] | 15360 [11695.6 to 20172.0] | 13663 [10498.8 to 17779.9] | 11805 [9135.4 to 15255.7] | 14570 [11447.8 to 18544.3] | 12273 [9077.2 to 16595.1] | 10764 [7824.2 to 14807.5] | 1718 [1389.8 to 2123.4]
  RSV A:6 Months after vaccination 1: number analyzed (Participants) | 37 | 37 | 40 | 38 | 38 | 39 | 38 | 35 | 38 | 38 | 40 | 36 | 38
  RSV A:6 Months after vaccination 1 | 8403 [6386.5 to 11056.6] | 8118 [6048.2 to 10896.6] | 9568 [7416.5 to 12343.6] | 9533 [7128.0 to 12748.9] | 6492 [4911.2 to 8580.7] | 10324 [7545.2 to 14125.7] | 10005 [7832.8 to 12780.0] | 10237 [7792.7 to 13447.1] | 7768 [5960.2 to 10123.8] | 10343 [7596.7 to 14082.5] | 8823 [6401.5 to 12160.3] | 8210 [5890.4 to 11443.8] | 2031 [1613.7 to 2556.1]
  RSV A: 12 Months after vaccination 1: number analyzed (Participants) | 34 | 36 | 37 | 33 | 36 | 36 | 33 | 33 | 37 | 36 | 33 | 31 | 32
  RSV A: 12 Months after vaccination 1 | 7679 [5830.0 to 10114.5] | 7050 [4686.3 to 10605.3] | 7640 [6033.3 to 9673.4] | 9062 [6616.6 to 12411.7] | 4889 [3243.0 to 7370.6] | 8435 [5784.9 to 12300.3] | 9174 [6766.8 to 12438.6] | 8231 [6167.4 to 10986.4] | 6919 [4936.1 to 9698.5] | 6983 [5099.0 to 9562.3] | 6769 [4811.0 to 9522.9] | 5658 [3602.1 to 8888.6] | 1994 [1445.8 to 2751.0]
  RSV B: before vaccination 1 | 1847 [1415.4 to 2410.9] | 1475 [1117.0 to 1949.1] | 1516 [1120.5 to 2050.8] | 1586 [1182.6 to 2127.6] | 1460 [1131.3 to 1884.3] | 1502 [1123.0 to 2010.2] | 1739 [1396.0 to 2166.4] | 1733 [1334.2 to 2251.6] | 1480 [1123.8 to 1949.5] | 1520 [1116.7 to 2067.9] | 1363 [1029.7 to 1803.0] | 1584 [1147.9 to 2185.8] | 1783 [1371.8 to 2316.9]
  RSV B: 1 Month after vaccination 1 | 17583 [13214.1 to 23395.6] | 19561 [15064.1 to 25399.1] | 18762 [13685.5 to 25721.9] | 16835 [12239.1 to 23157.8] | 18929 [14318.0 to 25025.3] | 24395 [18501.1 to 32165.3] | 23560 [18937.0 to 29311.1] | 22928 [16479.1 to 31901.0] | 23481 [17190.7 to 32072.3] | 31571 [25226.8 to 39511.5] | 21150 [15284.8 to 29265.8] | 28166 [21107.4 to 37585.2] | 1748 [1329.6 to 2299.0]
  RSV B: 2 Months after vaccination 1: number analyzed (Participants) | 38 | 38 | 39 | 38 | 39 | 39 | 39 | 35 | 40 | 39 | 39 | 38 | 41
  RSV B: 2 Months after vaccination 1 | 10259 [8034.9 to 13099.5] | 11771 [8638.2 to 16040.4] | 11441 [8386.4 to 15607.7] | 11253 [8111.2 to 15611.0] | 10486 [7919.2 to 13884.8] | 14223 [10536.4 to 19200.6] | 15173 [11310.1 to 20356.1] | 11716 [8515.6 to 16119.1] | 12850 [9187.3 to 17972.3] | 16485 [12365.4 to 21978.4] | 11148 [8237.5 to 15087.2] | 14024 [10061.6 to 19547.9] | 1447 [1079.9 to 1939.5]
  RSV B: 3 Months after vaccination 1: number analyzed (Participants) | 37 | 38 | 39 | 38 | 38 | 38 | 39 | 35 | 40 | 39 | 40 | 38 | 41
  RSV B: 3 Months after vaccination 1 | 11694 [8668.6 to 15774.1] | 12016 [9365.0 to 15416.8] | 12852 [9598.1 to 17209.5] | 11719 [8535.2 to 16091.6] | 9953 [7528.7 to 13159.2] | 13011 [9004.5 to 18800.0] | 13364 [10482.3 to 17038.8] | 11333 [8551.7 to 15018.5] | 10567 [8130.7 to 13732.8] | 14638 [11159.9 to 19200.0] | 10322 [7548.2 to 14113.9] | 11146 [7975.6 to 15576.6] | 1839 [1439.5 to 2349.4]
  RSV B: 6 Months after vaccination 1: number analyzed (Participants) | 37 | 37 | 40 | 38 | 38 | 39 | 38 | 35 | 38 | 38 | 40 | 36 | 38
  RSV B: 6 Months after vaccination 1 | 8102 [6262.1 to 10481.3] | 8411 [6558.5 to 10786.8] | 9954 [7389.7 to 13407.1] | 8667 [6315.1 to 11895.8] | 6640 [5134.2 to 8586.8] | 9482 [6798.6 to 13225.5] | 9702 [7732.8 to 12172.6] | 8836 [6541.4 to 11934.4] | 7244 [5597.4 to 9374.1] | 11073 [7984.1 to 15356.1] | 8235 [5889.9 to 11513.3] | 8856 [6341.0 to 12367.3] | 2171 [1687.8 to 2792.3]
  RSV B: 12 Months after vaccination 1: number analyzed (Participants) | 34 | 36 | 37 | 33 | 36 | 36 | 33 | 33 | 37 | 36 | 33 | 31 | 32
  RSV B: 12 Months after vaccination 1 | 7539 [5917.8 to 9603.1] | 7413 [5610.6 to 9795.7] | 7651 [5627.3 to 10403.5] | 7629 [5427.0 to 10723.6] | 5778 [4201.0 to 7947.8] | 7747 [5099.8 to 11767.6] | 8492 [6382.7 to 11297.8] | 7177 [5333.3 to 9658.8] | 6078 [4465.2 to 8274.7] | 7086 [5112.3 to 9820.9] | 6133 [4215.6 to 8923.1] | 5494 [3465.4 to 8710.7] | 2017 [1503.9 to 2705.9]

22. Secondary Outcome: Expanded Cohort: GMTs of RSV A and RSV B Antigens Following Vaccination in Participants (Aged 65 to 85 Years)
Description: as for outcome 20
Time Frame: Before vaccination, 1, 2, 3, 6 and 12 months after vaccination
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Number analyzed (Participants) | 38 | 40 | 40 | 40 | 38 | 40 | 40 | 40 | 40 | 38 | 41 | 43 | 39
Titers
  RSV A: before vaccination 1 | 2129 [1577.8 to 2872.8] | 2096 [1518.6 to 2892.0] | 2064 [1638.5 to 2598.9] | 2461 [1856.2 to 3262.5] | 2269 [1708.5 to 3013.4] | 2269 [1802.6 to 2855.8] | 2578 [1945.6 to 3416.6] | 2089 [1535.1 to 2843.5] | 2203 [1731.5 to 2802.0] | 1965 [1539.1 to 2508.5] | 1793 [1351.8 to 2378.8] | 2734 [1963.5 to 3807.4] | 1585 [1252.3 to 2005.5]
  RSV A: 1 Month after vaccination 1 | 16007 [12504.7 to 20489.7] | 20417 [14920.6 to 27937.5] | 14905 [11631.7 to 19098.2] | 19625 [14184.9 to 27151.3] | 25065 [19629.1 to 32006.7] | 22318 [15850.6 to 31425.6] | 23566 [17457.3 to 31812.3] | 27600 [21382.5 to 35624.6] | 22184 [16026.2 to 30708.8] | 21601 [16659.4 to 28007.6] | 23510 [17822.0 to 31013.3] | 25815 [19944.3 to 33412.8] | 1697 [1250.6 to 2301.8]
  RSV A: 2 Months after vaccination 1: number analyzed (Participants) | 38 | 40 | 40 | 40 | 38 | 40 | 39 | 40 | 40 | 38 | 41 | 43 | 39
  RSV A: 2 Months after vaccination 1 | 9452 [7428.7 to 12027.1] | 13199 [10283.1 to 16941.3] | 9922 [7222.7 to 13630.8] | 15484 [11526.9 to 20800.1] | 16288 [11911.8 to 22271.2] | 12740 [9523.2 to 17044.6] | 11939 [9013.1 to 15815.1] | 15840 [11770.4 to 21316.0] | 14438 [10978.8 to 18988.3] | 14542 [11233.0 to 18825.2] | 16797 [12172.8 to 23178.9] | 17410 [13396.9 to 22624.1] | 1414 [1074.8 to 1859.1]
  RSV A:3 Months after vaccination 1: number analyzed (Participants) | 36 | 40 | 40 | 39 | 38 | 39 | 39 | 39 | 40 | 38 | 41 | 43 | 39
  RSV A:3 Months after vaccination 1 | 12010 [9596.8 to 15028.9] | 14230 [10948.0 to 18497.1] | 10362 [7851.6 to 13675.7] | 15345 [11425.0 to 20610.2] | 16637 [13056.4 to 21199.4] | 14957 [11432.2 to 19567.5] | 13675 [9813.9 to 19056.4] | 16424 [12590.9 to 21424.4] | 16089 [12483.9 to 20735.6] | 12200 [9656.1 to 15413.8] | 15291 [11066.0 to 21130.2] | 16265 [12538.4 to 21100.0] | 1772 [1437.1 to 2185.9]
  RSV A:6 Months after vaccination 1: number analyzed (Participants) | 38 | 40 | 40 | 39 | 38 | 40 | 39 | 39 | 40 | 38 | 41 | 43 | 38
  RSV A:6 Months after vaccination 1 | 8452 [6630.3 to 10775.1] | 11903 [9294.4 to 15242.5] | 8444 [6262.1 to 11385.4] | 10827 [8198.8 to 14299.0] | 11871 [8636.7 to 16317.0] | 10202 [7456.7 to 13958.5] | 10226 [7555.1 to 13840.9] | 13148 [10485.1 to 16487.1] | 10769 [8228.7 to 14092.3] | 9495 [7587.8 to 11881.8] | 10578 [7678.5 to 14571.9] | 11268 [8581.1 to 14795.8] | 2057 [1480.4 to 2859.3]
  RSV A: 12 Months after vaccination 1: number analyzed (Participants) | 38 | 39 | 40 | 37 | 36 | 40 | 38 | 36 | 37 | 36 | 41 | 43 | 38
  RSV A: 12 Months after vaccination 1 | 7732 [5994.9 to 9971.5] | 7891 [5743.4 to 10841.2] | 6518 [4825.7 to 8804.0] | 9143 [6587.4 to 12689.9] | 7942 [4956.1 to 12728.1] | 8639 [6159.4 to 12116.2] | 7731 [5491.0 to 10885.4] | 9340 [6921.2 to 12603.7] | 9738 [7079.7 to 13394.9] | 5872 [3775.9 to 9132.2] | 6946 [4590.1 to 10510.8] | 8919 [6166.3 to 12899.3] | 1931 [1440.0 to 2590.3]
  RSV B: before vaccination 1: number analyzed (Participants) | 38 | 40 | 40 | 40 | 38 | 40 | 40 | 39 | 40 | 38 | 41 | 43 | 39
  RSV B: before vaccination 1 | 2198 [1573.7 to 3070.9] | 1862 [1340.9 to 2586.5] | 1999 [1506.1 to 2653.9] | 2423 [1840.0 to 3191.1] | 2314 [1659.8 to 3225.1] | 2194 [1724.9 to 2790.8] | 2685 [1949.1 to 3698.5] | 2032 [1414.4 to 2920.4] | 2586 [1999.1 to 3344.0] | 2241 [1689.0 to 2972.7] | 1635 [1155.3 to 2313.4] | 2390 [1744.5 to 3274.4] | 1766 [1371.2 to 2275.6]
  RSV B: 1 Month after vaccination 1 | 15172 [10995.0 to 20936.5] | 20553 [14241.6 to 29660.2] | 15169 [11469.2 to 20063.1] | 20421 [13852.5 to 30105.7] | 24257 [17639.8 to 33356.3] | 18648 [12034.5 to 28896.9] | 24158 [16688.4 to 34969.9] | 30071 [21347.9 to 42359.2] | 27996 [19063.0 to 41115.9] | 25080 [17447.2 to 36052.5] | 24320 [17529.7 to 33741.2] | 25719 [18637.2 to 35491.1] | 1664 [1229.2 to 2252.4]
  RSV B: 2 Months after vaccination 1: number analyzed (Participants) | 38 | 40 | 40 | 40 | 38 | 40 | 39 | 40 | 40 | 38 | 41 | 43 | 39
  RSV B: 2 Months after vaccination 1 | 9162 [6658.1 to 12608.1] | 14085 [10386.5 to 19100.9] | 9928 [6957.8 to 14166.3] | 16107 [11164.1 to 23237.5] | 14496 [9907.2 to 21210.5] | 10893 [7861.3 to 15092.6] | 11605 [8207.0 to 16410.6] | 17024 [11790.9 to 24580.3] | 17255 [12641.8 to 23552.0] | 16376 [11778.6 to 22767.4] | 17706 [12608.5 to 24864.7] | 17268 [13010.8 to 22917.7] | 1413 [1093.7 to 1824.7]
  RSV B: 3 Months after vaccination 1: number analyzed (Participants) | 36 | 40 | 40 | 39 | 38 | 39 | 39 | 39 | 40 | 38 | 41 | 43 | 39
  RSV B: 3 Months after vaccination 1 | 12578 [8794.3 to 17989.3] | 13735 [10112.3 to 18654.7] | 9741 [6327.5 to 14996.3] | 15856 [11221.3 to 22404.0] | 14163 [10608.8 to 18908.1] | 11927 [8704.5 to 16343.6] | 13631 [9258.0 to 20070.2] | 16675 [11847.7 to 23468.8] | 18557 [13406.8 to 25686.3] | 13452 [9659.9 to 18731.6] | 15031 [10537.4 to 21442.2] | 14645 [10736.8 to 19976.6] | 1995 [1627.0 to 2446.5]
  RSV B: 6 Months after vaccination 1: number analyzed (Participants) | 38 | 40 | 40 | 39 | 38 | 40 | 39 | 39 | 40 | 38 | 41 | 43 | 38
  RSV B: 6 Months after vaccination 1 | 8429 [6127.1 to 11596.0] | 11417 [8472.7 to 15384.7] | 7869 [5884.7 to 10521.8] | 11739 [8330.6 to 16542.4] | 10606 [7585.3 to 14830.1] | 9270 [6321.4 to 13592.7] | 10384 [6793.2 to 15872.9] | 13562 [10077.8 to 18251.6] | 11710 [8535.9 to 16064.2] | 10597 [7911.2 to 14195.9] | 10645 [7424.7 to 15262.1] | 10875 [8159.0 to 14496.1] | 2374 [1633.3 to 3452.0]
  RSV B: 12 Months after vaccination 1: number analyzed (Participants) | 38 | 39 | 40 | 37 | 36 | 40 | 38 | 36 | 37 | 36 | 41 | 43 | 38
  RSV B: 12 Months after vaccination 1 | 7467 [5426.5 to 10274.0] | 7969 [5671.5 to 11196.5] | 6445 [4561.6 to 9106.0] | 9200 [6460.4 to 13101.5] | 7573 [4659.2 to 12310.2] | 6634 [4565.5 to 9639.4] | 7449 [5139.4 to 10796.7] | 9256 [6496.9 to 13186.5] | 9855 [6874.6 to 14127.4] | 6809 [4274.8 to 10846.9] | 7001 [4436.2 to 11049.8] | 8500 [5551.2 to 13016.2] | 2058 [1525.8 to 2775.8]

23. Secondary Outcome: Expanded Cohort: Hemagglutination Inhibition Assay (HAI) Titers for All Strains Following Vaccination With Seasonal Inactivated Influenza (SIIV) Vaccine in Participants (Aged 18 to 49 Years)
Description: The HAI titer LLOQ value for each strain was 10. Assay values below LLOQ were set to 0.5* LLOQ for analysis. Titers were expressed in terms of 1/dilution.
Time Frame: Before vaccination and 1 Month after SIIV vaccination
Population: Evaluable influenza immunogenicity population (EIIP) : participants who were eligible, received all RSV vaccine or placebo to which they were randomized, received influenza vaccine, had blood drawn for assay testing within 27 to 42 days after Visit 1, had at least 1 valid and determinate assay result at 1-month-postvaccination visit and no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years
Number analyzed (Participants) | 39 | 33 | 40 | 32 | 40 | 33 | 39 | 33 | 40 | 36 | 41 | 31 | 34
Titers
  A-H1N1: before SIIV | 44.5 [30.34 to 65.26] | 25.0 [17.15 to 36.51] | 38.0 [25.74 to 56.03] | 33.7 [22.47 to 50.53] | 18.9 [13.51 to 26.47] | 27.0 [16.99 to 42.96] | 29.6 [19.01 to 45.99] | 26.1 [16.68 to 40.85] | 20.5 [14.21 to 29.48] | 28.7 [18.16 to 45.28] | 32.1 [22.97 to 44.88] | 22.7 [14.61 to 35.35] | 33.5 [21.85 to 51.43]
  A-H1N1: 1 month after SIIV | 77.2 [55.13 to 108.07] | 95.3 [65.73 to 138.06] | 85.8 [63.75 to 115.37] | 114.0 [75.09 to 173.00] | 62.4 [45.56 to 85.46] | 113.5 [73.56 to 175.25] | 70.2 [46.13 to 106.88] | 128.8 [87.91 to 188.58] | 57.2 [43.42 to 75.40] | 83.6 [58.45 to 119.71] | 72.3 [54.40 to 96.16] | 114.4 [81.16 to 161.24] | 126.9 [91.78 to 175.60]
  A-H3N2: before SIIV | 35.1 [23.42 to 52.58] | 25.4 [16.15 to 39.89] | 32.7 [22.27 to 47.91] | 35.7 [22.14 to 57.44] | 23.9 [15.90 to 36.02] | 28.8 [18.02 to 45.95] | 30.3 [18.90 to 48.56] | 25.7 [15.10 to 43.83] | 20.9 [13.37 to 32.81] | 22.4 [14.54 to 34.63] | 32.3 [21.51 to 48.44] | 20.3 [13.25 to 31.06] | 34.4 [23.03 to 51.44]
  A-H3N2: 1 month after SIIV | 77.7 [54.76 to 110.11] | 129.6 [84.87 to 198.00] | 81.4 [58.32 to 113.57] | 158.8 [113.23 to 222.77] | 85.2 [57.22 to 126.96] | 120.0 [77.87 to 185.00] | 74.5 [50.39 to 110.25] | 130.6 [83.11 to 205.23] | 81.4 [59.53 to 111.30] | 82.1 [56.50 to 119.19] | 95.8 [67.10 to 136.84] | 134.8 [92.88 to 195.69] | 152.5 [114.26 to 203.64]
  B1: before SIIV | 13.2 [9.24 to 18.73] | 10.3 [7.64 to 13.87] | 10.8 [7.81 to 14.93] | 13.3 [8.97 to 19.86] | 7.3 [5.92 to 9.06] | 13.0 [9.12 to 18.43] | 8.7 [6.61 to 11.53] | 9.5 [6.64 to 13.46] | 8.3 [6.27 to 11.03] | 9.4 [6.75 to 13.22] | 12.6 [9.30 to 17.06] | 9.2 [6.77 to 12.55] | 10.5 [8.05 to 13.68]
  B1: 1 month after SIIV | 23.5 [17.09 to 32.25] | 41.7 [27.86 to 62.52] | 29.3 [20.47 to 41.97] | 47.2 [29.73 to 74.99] | 18.4 [13.75 to 24.74] | 38.4 [25.91 to 56.86] | 19.1 [13.83 to 26.41] | 32.7 [20.81 to 51.27] | 15.5 [11.28 to 21.39] | 22.3 [15.61 to 31.85] | 23.8 [18.32 to 30.95] | 25.6 [16.86 to 38.82] | 31.8 [21.21 to 47.55]
  B2: before SIIV | 16.3 [11.09 to 23.85] | 11.7 [8.93 to 15.24] | 12.5 [9.29 to 16.71] | 18.4 [12.60 to 26.73] | 9.3 [7.16 to 12.20] | 12.8 [9.20 to 17.77] | 11.5 [8.68 to 15.30] | 10.6 [7.32 to 15.27] | 10.4 [7.84 to 13.83] | 12.3 [8.75 to 17.25] | 11.6 [8.73 to 15.53] | 11.2 [8.19 to 15.31] | 13.1 [9.74 to 17.69]
  B2: 1 month after SIIV | 29.0 [21.07 to 40.04] | 39.4 [27.06 to 57.46] | 27.8 [20.40 to 37.97] | 46.9 [31.34 to 70.31] | 22.6 [17.56 to 29.11] | 28.4 [18.66 to 43.17] | 22.3 [16.17 to 30.65] | 39.7 [25.21 to 62.56] | 20.1 [14.73 to 27.51] | 28.7 [20.16 to 40.71] | 25.9 [19.08 to 35.19] | 37.5 [27.37 to 51.25] | 36.2 [26.26 to 49.80]

24. Secondary Outcome: Expanded Cohort: Hemagglutination Inhibition Assay (HAI) Titers for All Strains Following Vaccination With Seasonal Inactivated Influenza (SIIV) Vaccine in Participants (Aged 65 to 85 Years)
Description: as for outcome 23
Time Frame: Before vaccination and 1 Month after SIIV vaccination
Population: EIIP : participants who were eligible, received all RSV vaccine or placebo to which they were randomized, received influenza vaccine, had blood drawn for assay testing within 27 to 42 days after Visit 1, had at least 1 valid and determinate assay result at 1-month-postvaccination visit and no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
Number analyzed (Participants) | 38 | 35 | 40 | 36 | 38 | 37 | 40 | 37 | 40 | 33 | 41 | 35 | 34
Titers
  A-H1N1: before SIIV | 13.8 [10.12 to 18.94] | 14.8 [9.94 to 21.93] | 11.0 [8.67 to 13.87] | 13.4 [9.34 to 19.10] | 16.6 [11.42 to 24.03] | 12.3 [8.63 to 17.53] | 17.5 [11.91 to 25.74] | 14.4 [10.84 to 19.26] | 17.8 [12.69 to 25.00] | 15.2 [11.37 to 20.39] | 15.6 [11.14 to 21.87] | 22.5 [14.87 to 34.10] | 17.6 [11.89 to 26.00]
  A-H1N1: 1 month after SIIV | 43.6 [29.44 to 64.44] | 54.5 [36.01 to 82.60] | 44.4 [30.05 to 65.55] | 61.9 [44.30 to 86.50] | 52.9 [37.69 to 74.31] | 51.1 [33.92 to 76.97] | 56.6 [36.12 to 88.61] | 71.0 [50.60 to 99.77] | 45.7 [31.63 to 66.00] | 58.4 [40.56 to 84.11] | 52.4 [33.76 to 81.37] | 72.0 [48.76 to 106.23] | 75.8 [52.94 to 108.40]
  A-H3N2: before SIIV | 29.7 [20.41 to 43.23] | 24.7 [16.39 to 37.24] | 26.2 [16.56 to 41.58] | 22.9 [14.25 to 36.72] | 34.6 [21.08 to 56.69] | 23.5 [16.45 to 33.66] | 30.5 [19.70 to 47.20] | 35.7 [20.99 to 60.84] | 22.5 [14.37 to 35.11] | 32.6 [21.12 to 50.40] | 34.7 [21.82 to 55.29] | 44.5 [28.03 to 70.66] | 28.7 [17.54 to 46.87]
  A-H3N2: 1 month after SIIV | 94.3 [62.80 to 141.58] | 105.6 [67.56 to 164.96] | 78.2 [50.07 to 122.27] | 118.3 [78.75 to 177.68] | 140.0 [95.48 to 205.23] | 109.3 [69.69 to 171.51] | 131.5 [87.38 to 197.83] | 185.0 [107.84 to 317.50] | 79.0 [55.60 to 112.38] | 153.4 [98.53 to 238.89] | 103.1 [63.41 to 167.73] | 130.4 [76.49 to 222.29] | 106.4 [64.27 to 176.25]
  B1: before SIIV | 9.4 [6.86 to 12.77] | 8.6 [6.40 to 11.56] | 12.9 [8.78 to 18.95] | 8.5 [6.73 to 10.79] | 11.1 [7.96 to 15.47] | 10.4 [7.56 to 14.26] | 11.5 [8.26 to 15.97] | 8.7 [6.61 to 11.37] | 8.7 [6.69 to 11.34] | 8.5 [6.56 to 10.91] | 9.5 [6.97 to 12.97] | 8.6 [6.56 to 11.39] | 9.1 [7.08 to 11.67]
  B1: 1 month after SIIV | 19.5 [13.45 to 28.32] | 26.4 [17.77 to 39.22] | 22.9 [16.22 to 32.19] | 31.7 [22.89 to 43.96] | 24.7 [16.82 to 36.39] | 23.4 [16.25 to 33.69] | 26.2 [17.56 to 39.20] | 21.6 [15.13 to 30.72] | 18.9 [12.77 to 27.89] | 29.4 [19.44 to 44.45] | 21.2 [15.17 to 29.64] | 23.1 [16.58 to 32.32] | 26.8 [17.35 to 41.34]
  B2: before SIIV | 7.7 [6.19 to 9.46] | 7.7 [6.16 to 9.58] | 9.6 [7.26 to 12.72] | 8.0 [6.24 to 10.23] | 10.6 [7.55 to 14.99] | 8.2 [6.24 to 10.75] | 9.9 [7.37 to 13.25] | 6.9 [5.60 to 8.45] | 7.9 [6.21 to 10.15] | 8.3 [6.69 to 10.26] | 8.6 [6.66 to 11.10] | 8.4 [6.88 to 10.33] | 7.3 [5.71 to 9.38]
  B2: 1 month after SIIV | 10.4 [8.00 to 13.44] | 11.0 [8.01 to 15.02] | 13.0 [9.15 to 18.37] | 12.4 [8.84 to 17.30] | 16.6 [11.67 to 23.50] | 13.2 [9.48 to 18.31] | 13.3 [9.49 to 18.76] | 10.0 [7.94 to 12.62] | 9.7 [7.57 to 12.35] | 15.3 [10.49 to 22.39] | 10.9 [8.02 to 14.77] | 13.2 [9.99 to 17.46] | 13.2 [9.13 to 19.16]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events collected as Non-SAEs: within 14 days after Vaccination (Vax) 1 and Vax 3 (for revaccination); Other Non-SAEs: Vax 1 up to 1 month after Vax 1, Vax 3 up to 1 month after Vax 3 for revaccination; SAEs: Vax 1 up to 12 months after Vax 1 (approximately up to 378 days), Vax 1 up to 12 months after Vax 3 for revaccination (approximately up to 798 days)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Groups:
- Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years:: Participants aged 18-49 years received RSV vaccine 120 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years: Participants aged 18-49 years received RSV vaccine 60 mcg along with aluminum hydroxide and 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years:: Participants aged 65-85 years received RSV vaccine 120 mcg along with 0.5 mL SIIV intramuscularly at Day 1 (Vaccination 1). Participants received placebo (saline control) intramuscularly at Day 35 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
Arm/Group | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years | Sentinel Cohort: RSV 120 mcg Age 18-49 Years | Sentinel Cohort: RSV 240 mcg Age 18-49 Years | Sentinel Cohort: Placebo Age 18-49 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years | Sentinel Cohort: RSV 120 mcg Age 50-85 Years | Sentinel Cohort: RSV 240 mcg Age 50-85 Years | Sentinel Cohort: Placebo Age 50-85 Years | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years: | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years: | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 1/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/41 | 0/41 | 0/41 | 0/41 | 1/41 | 0/41 | 0/41 | 0/41 | 0/42 | 0/40 | 1/41 | 1/41 | 0/43 | 0/42 | 0/40 | 1/41 | 0/41 | 0/41 | 0/41 | 0/40 | 0/40 | 0/40 | 1/41 | 0/40 | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 2/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 1/12 | 0/12 | 1/41 | 0/41 | 1/41 | 0/41 | 2/41 | 1/41 | 2/41 | 7/41 | 8/42 | 2/40 | 2/41 | 5/41 | 3/43 | 0/42 | 1/40 | 2/41 | 2/41 | 3/41 | 3/41 | 2/40 | 4/40 | 4/40 | 7/41 | 5/40 | 4/42 | 3/41
Other Adverse Events (participants affected / at risk) | 9/12 | 6/12 | 7/12 | 6/12 | 7/12 | 7/12 | 8/12 | 10/12 | 11/12 | 9/12 | 8/12 | 5/12 | 5/12 | 4/12 | 31/41 | 36/41 | 33/41 | 35/41 | 35/41 | 35/41 | 31/41 | 24/41 | 27/42 | 22/40 | 25/41 | 28/41 | 33/43 | 32/42 | 30/40 | 33/41 | 35/41 | 32/41 | 38/41 | 22/40 | 20/40 | 21/40 | 21/41 | 32/40 | 29/42 | 21/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years (N=12) | Sentinel Cohort: RSV 120 mcg Age 18-49 Years (N=12) | Sentinel Cohort: RSV 240 mcg Age 18-49 Years (N=12) | Sentinel Cohort: Placebo Age 18-49 Years (N=12) | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years (N=12) | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years (N=12) | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years (N=12) | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years (N=12) | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years (N=12) | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years (N=12) | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years (N=12) | Sentinel Cohort: RSV 120 mcg Age 50-85 Years (N=12) | Sentinel Cohort: RSV 240 mcg Age 50-85 Years (N=12) | Sentinel Cohort: Placebo Age 50-85 Years (N=12) | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years: (N=41) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years (N=41) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years (N=42) | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years (N=40) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years (N=41) | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years (N=41) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years (N=43) | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years (N=42) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years (N=40) | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years (N=40) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years (N=40) | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years: (N=40) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years (N=41) | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years (N=40) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years (N=42) | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Maisonneuve fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autonomic failure syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy of partner (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Sentinel Cohort: RSV Vaccine 60 mcg Age 18-49 Years (N=12) | Sentinel Cohort: RSV 120 mcg Age 18-49 Years (N=12) | Sentinel Cohort: RSV 240 mcg Age 18-49 Years (N=12) | Sentinel Cohort: Placebo Age 18-49 Years (N=12) | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 50-85 Years (N=12) | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 50-85 Years (N=12) | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 50-85 Years (N=12) | Sentinel Cohort: RSV 60 mcg With Aluminum Hydroxide Age 18-49 Years (N=12) | Sentinel Cohort: RSV 120 mcg With Aluminum Hydroxide Age 18-49 Years (N=12) | Sentinel Cohort: RSV 240 mcg With Aluminum Hydroxide Age 18-49 Years (N=12) | Sentinel Cohort: RSV Vaccine 60 mcg Age 50-85 Years (N=12) | Sentinel Cohort: RSV 120 mcg Age 50-85 Years (N=12) | Sentinel Cohort: RSV 240 mcg Age 50-85 Years (N=12) | Sentinel Cohort: Placebo Age 50-85 Years (N=12) | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 18-49 Years: (N=41) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 18-49 Years (N=41) | Expanded Cohort: Placebo and Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 65-85 Years (N=41) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years (N=42) | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 65-85 Years (N=40) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years (N=41) | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 65-85 Years (N=41) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 65-85 Years (N=43) | Expanded Cohort: RSV 60 mcg With Placebo and SIIV Age 18-49 Years (N=42) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years (N=40) | Expanded Cohort: RSV 120 mcg With Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and Placebo and SIIV Age 18-49 Years (N=41) | Expanded Cohort: RSV 60 mcg With SIIV and Placebo Age 65-85 Years (N=40) | Expanded Cohort: RSV 60 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years (N=40) | Expanded Cohort: RSV 120 mcg With SIIV and Placebo Age 65-85 Years: (N=40) | Expanded Cohort: RSV 120 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years (N=41) | Expanded Cohort: RSV 240 mcg With SIIV and Placebo Age 65-85 Years (N=40) | Expanded Cohort: RSV 240 mcg With Aluminum Hydroxide and SIIV and Placebo Age 65-85 Years (N=42) | Expanded Cohort: Placebo and Placebo and SIIV Age 65-85 Years (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (REDNESS) (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 3 | 4 | 1 | 2/40 | 4 | 3 | 1 | 6 | 3 | 3 | 1 | 2 | 3/40 | 2 | 6 | 3 | 1 | 3 | 2 | 2 | 1 | 0/40 — 11 participants of sentinel cohort:RSV 240 mcg age 18-49 years,40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 years,RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) arms were at risk.
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site pain (PAIN AT INJECTION SITE) (General disorders) | 6 | 3 | 2/11 | 2 | 3 | 5 | 2 | 9 | 10 | 8 | 2 | 1 | 1 | 0 | 19 | 28 | 19 | 25 | 27 | 30 | 10 | 4/40 | 10 | 5 | 8 | 16 | 16 | 16 | 21 | 21 | 27/40 | 24 | 30 | 11 | 11 | 9 | 12 | 17 | 17 | 2/40 — 11 participants of sentinel cohort:RSV 240 mcg age 18-49 years,40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 years,RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) arms were at risk.
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site swelling (SWELLING) (General disorders) | 0 | 0 | 0/11 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 5 | 4 | 0 | 2/40 | 2 | 2 | 1 | 4 | 5 | 4 | 1 | 4 | 2/40 | 2 | 10 | 3 | 0 | 3 | 1 | 4 | 5 | 1/40 — 11 participants of sentinel cohort:RSV 240 mcg age 18-49 years,40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 years,RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) arms were at risk.
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (FEVER) (General disorders) | 0 | 0 | 0/11 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 2 | 0 | 0 | 1/40 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 2 | 0/40 | 2 | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 0/40 — 11 participants of sentinel cohort:RSV 240 mcg age 18-49 years,40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 years,RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) arms were at risk
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 1 | 2 | 3/11 | 1 | 0 | 1 | 2 | 3 | 2 | 1 | 0 | 2 | 4 | 1 | 6 | 10 | 10 | 8 | 11 | 9 | 6 | 7/40 | 5 | 2 | 6 | 5 | 7 | 10 | 7 | 10 | 10/40 | 11 | 14 | 3 | 9 | 4 | 4 | 10 | 8 | 6/40 — 11 participants(sentinel cohort:RSV 240 mcg age 18-49 years arm),40 participants(expanded cohort:RSV 120 mcg with aluminum hydroxide and placebo and SIIV Age 18-49 Years arm)40 participants for placebo & placebo & SIIV Age 65-85 years were at risk.
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 3 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 3 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure systolic decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2/11 | 1 | 4 | 4 | 2 | 1 | 2 | 2 | 2 | 0 | 1 | 1 | 8 | 11 | 8 | 10 | 11 | 9 | 5 | 7/40 | 8 | 6 | 8 | 7 | 6 | 5 | 2 | 5 | 12/40 | 11 | 9 | 8 | 4 | 6 | 5 | 6 | 14 | 7/40 — 11 participants of sentinel cohort: RSV 240 mcg age 18-49 years, 40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 Years, RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) were at risk.
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 6 | 4 | 2/11 | 1 | 4 | 6 | 4 | 4 | 6 | 7 | 4 | 1 | 2 | 1 | 17 | 23 | 14 | 25 | 19 | 23 | 9 | 6/40 | 7 | 5 | 11 | 16 | 11 | 13 | 15 | 17 | 21/40 | 19 | 26 | 7 | 6 | 9 | 8 | 18 | 18 | 5/40 — 11 participants of sentinel cohort: RSV 240 mcg age 18-49 years, 40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 Years, RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) were at risk.
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (FATIGUE) (General disorders) | 5 | 5 | 6/11 | 3 | 7 | 4 | 3 | 6 | 7 | 7 | 5 | 4 | 1 | 4 | 20 | 17 | 16 | 18 | 21 | 24 | 18 | 10/40 | 16 | 8 | 13 | 12 | 16 | 19 | 16 | 15 | 20/40 | 25 | 20 | 8 | 11 | 9 | 14 | 20 | 21 | 8/40 — 11 participants of sentinel cohort: RSV 240 mcg age 18-49 years, 40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 Years, RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) were at risk.
Nausea (NAUSEA) (Gastrointestinal disorders) | 4 | 2 | 2/11 | 0 | 1 | 1 | 2 | 0 | 2 | 3 | 2 | 2 | 1 | 0 | 6 | 8 | 6 | 5 | 12 | 4 | 8 | 4/40 | 1 | 2 | 8 | 6 | 3 | 6 | 6 | 11 | 9/40 | 7 | 10 | 2 | 1 | 2 | 4 | 7 | 5 | 3/40 — 11 participants(sentinel cohort)RSV 240 mcg age 18-49 years,40 participants(expanded cohort)RSV 120 mcg with aluminum hydroxide &placebo&SIIV age18-49 Years&40 participants(expanded cohort) placebo & placebo & SIIV Age 65-85 Years arms were at risk.
Vomiting (VOMITING) (Gastrointestinal disorders) | 1 | 0 | 2/11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 3 | 1 | 2/40 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 1/40 | 1 | 4 | 0 | 0 | 0 | 0 | 2 | 0 | 1/40 — 11 participant of sentinel cohort: RSV 240 mcg age 18-49 years arm, 40 participants of expanded cohort: RSV 120 mcg with Al(OH)3 and placebo age 18-49 years and 40 participants of expanded Cohort: placebo age 65-85 years arms were at risk.
Headache (HEADACHE) (Nervous system disorders) | 5 | 3 | 7/11 | 1 | 3 | 3 | 1 | 5 | 5 | 5 | 1 | 1 | 3 | 1 | 18 | 16 | 21 | 19 | 26 | 21 | 17 | 5/40 | 7 | 7 | 10 | 12 | 16 | 23 | 18 | 20 | 19/40 | 19 | 20 | 10 | 5 | 7 | 4 | 11 | 15 | 10/40 — 11 participants of sentinel cohort: RSV 240 mcg age 18-49 years, 40 participants of expanded cohort (RSV 120 mcg with aluminum hydroxide and placebo age 18-49 Years, RSV 60 mcg with placebo age 65-85 years and placebo age 65-85 years) were at risk.
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03529773/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03529773/SAP_001.pdf